CLINICAL TRIAL: NCT01815424
Title: A PHASE 3, MULTI SITE, RANDOMIZED, DOUBLE BLIND, PLACEBO CONTROLLED, PARALLEL-GROUP STUDY OF THE EFFICACY AND SAFETY OF 2 ORAL DOSES OF CP-690,550 IN ASIAN SUBJECTS WITH MODERATE TO SEVERE CHRONIC PLAQUE PSORIASIS
Brief Title: A Study Evaluating The Efficacy And Safety Of CP-690,550 In Asian Subjects With Moderate To Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921174
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis
Keywords: Tofacitinib; CP-690; 550; Xeljanz; Jak-Inhibitor; Oral Treatment; Psoriasis vulgaris; Pruritus; Itch; DLQI; moderate; severe; chronic; plaque psoriasis
MeSH Terms: conditions — Psoriasis; Pruritus; Lymphoma, Follicular; Bronchiolitis Obliterans Syndrome | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo BID (Placebo Comparator)
  Interventions: Drug: placebo
- 5mg BID CP-690,550 (Experimental)
  Interventions: Drug: CP-690,550
- 10mg BID CP-690,550 (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: placebo — placebo BID for 16 weeks and then re-randomized into active groups
  Arms: Placebo BID
Drug: CP-690,550 — CP-690,550 5mg BID for 52 weeks
  Arms: 5mg BID CP-690,550
Drug: CP-690,550 — CP-690,550 10mg BID for 52 weeks
  Arms: 10mg BID CP-690,550

SUMMARY:
The primary objective of this study is to compare the efficacy of CP-690,550 (5 mg BID and 10 mg BID) versus placebo for the reduction in severity of plaque psoriasis after 16 weeks of treatment in Asian subjects with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of plaque-type psoriasis (psoriasis vulgaris) for at least 12 months prior to the first screening procedure.
* Have a PASI score of 12 or greater AND a PGA score of 3 ("moderate") or 4 ("severe") at Baseline (Day 1).
* Considered by dermatologist investigator to be a candidate for systemic therapy or phototherapy of psoriasis (either naïve or history of previous treatment).

Exclusion Criteria:

* Currently have non-plaque forms of psoriasis, eg, erythrodermic, guttate, or pustular psoriasis, with the exception of nail psoriasis which is allowed.
* Have current drug induced psoriasis, eg, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, antimalarial drugs or lithium.
* Subjects who cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot discontinue phototherapy (UVB or PUVA) for the study are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- China (18):
  - Dept. Of dermatology &STD, Beijing Friendship Hospital, Capital Medical University, Xicheng District, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hospital of Skin Diseases, Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Department of Dermatology, The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Huashan Hospital, Fudan University/Dermatology Department, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Dermatology Department, Shanghai, Shanghai Municipality
  - Dermatology Department, The First Affiliated Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of College of Medicine, Zhejiang University/Dermatology and STD Dept, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Peking University First Hospital / The Department of Dermatology, Beijing
  - Peking University People's Hospital/Dermatology Department, Beijing
  - Beijing Hospital of the Ministry of Health/Department of Dermatology, Beijing
  - Peking Union Medical College Hospital/Department of Dermatology, Beijing
  - Tianjin Medical University General Hospital, Dermatological Department, Tianjin
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Department of Dermatology,Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (3):
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Zhang J, Tsai TF, Lee MG, Zheng M, Wang G, Jin H, Gu J, Li R, Liu Q, Chen J, Tu C, Qi C, Zhu H, Ports WC, Crook T. The efficacy and safety of tofacitinib in Asian patients with moderate to severe chronic plaque psoriasis: A Phase 3, randomized, double-blind, placebo-controlled study. J Dermatol Sci. 2017 Oct;88(1):36-45. doi: 10.1016/j.jdermsci.2017.05.004. Epub 2017 May 16. PMID 28558978
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921174&StudyName=A%20Study%20Evaluating%20The%20Efficacy%20And%20Safety%20oO%20CP-690%2C550%20In%20Asian%20Subjects%20With%20Moderate%20To%20Severe%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib 10 mg: Participants received tofacitinib 10 mg tablet orally twice daily (approximately 12 hours apart) up to Week 52.
- Tofacitinib 5 mg: Participants received tofacitinib 5 mg tablet orally twice daily (approximately 12 hours apart) up to Week 52.
- Placebo: Participants received placebo tablets orally twice daily up to Week 16. At Week 16, participants in this group were automatically advanced to their second treatment of tofacitinib 5 mg or 10 mg tablet orally twice daily, which was pre-determined at randomization (44 participants assigned to Placebo to 5 mg, 44 participants assigned to Placebo to 10 mg).
- Placebo to Tofacitinib 10 mg: Participants received placebo tablet orally twice daily until Week 16, followed by tofacitinib 10 mg twice daily up to Week 52.
- Placebo to Tofacitinib 5 mg: Participants received placebo tablet orally twice daily until Week 16, followed by tofacitinib 5 mg twice daily up to Week 52.
Period: Week 0 to 16
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Started | 90 | 88 | 88 | 0 | 0
Completed | 83 | 84 | 77 | 0 | 0
Not Completed | 7 | 4 | 11 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 3 | 0 | 0
Not completed — Does Not Meet Entrance Criteria | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Insufficient Clinical Response | 2 | 0 | 4 | 0 | 0
Period: Week 16 to 52
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Started | 83 | 84 | 0 | 38 | 39
Completed | 81 | 79 | 0 | 35 | 36
Not Completed | 2 | 5 | 0 | 3 | 3
Not completed — Other | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Insufficient Clinical Response | 1 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis population included all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo | Total
Number analyzed (Participants) | 90 | 88 | 88 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.0) | 40.7 (11.3) | 41.7 (13.7) | 41.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 26 | 72
  Male | 67 | 65 | 62 | 194

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Physician's Global Assessment (PGA) Score of "Clear" or "Almost Clear" at Week 16
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear).
Time Frame: Week 16
Population: The full analysis population included all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo. Non-Responder Imputation (NRI) method (participants with missing values considered as non-responders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
percentage of participants | 75.56 | 52.27 | 19.32
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; For primary endpoint, step-down procedure used to preserve Type I error, sequential order of testing: PGA response for tofacitinib 10 mg vs placebo at Week 16; PASI75 response for tofacitinib 10 mg vs placebo at Week 16; PGA response for tofacitinib 5 mg vs placebo at Week 16; PASI75 response for tofacitinib 5 mg vs placebo at Week 16. If comparison at preceding step was significant, only then subsequent comparison was tested at the below specified significance level; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel statistics adjusted for pooled investigator sites was used for the analysis. Each hypothesis was tested at a significance level of 0.05 (2-sided); Odds Ratio (OR) = 14.52, 95% CI 2-sided [6.03 to 32.77]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.27, 95% CI 2-sided [2.46 to 11.86]

2. Primary Outcome: Percentage of Participants Achieving at Least a 75% Reduction in PASI (PASI75) at Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least a 75% reduction in PASI relative to Baseline.
Time Frame: Week 16
Population: The full analysis population included all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo. NRI method (participants with missing values considered as non-responders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
percentage of participants | 81.11 | 54.55 | 12.50
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 41.71, 95% CI 2-sided [14.84 to 151.11]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 9.97, 95% CI 2-sided [4.06 to 25.17]

3. Secondary Outcome: Percent Change From Baseline in Total Body Surface Area (BSA) With Psoriasis at Week 16
Description: Assessment of BSA with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints with percentage [Head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), Trunk (including axillae and groin) = 30% (30 handprints), lower extremities (including buttocks) = 40% (40 handprints)]. The number of handprints of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis. The total BSA affected was the summation of individual regions affected.
Time Frame: Baseline to Week 16
Population: The full analysis population included all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo. Number of participants analyzed was the evaluable participants for the specific criteria.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 84 | 84 | 77
percent change | -73.81 (5.903) | -54.39 (5.838) | -2.27 (6.061)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; This is a key secondary endpoint; family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant, only then subsequent comparison was tested at the below specified significance level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed model with fixed effects for treatment, visit, treatment-by-visit interaction, baseline value, and a random effect of subject; unstructured covariance matrix was used. Each hypothesis was tested at a significance of 0.025 (2-sided); Least Square Mean Difference = -71.54, 95% CI 2-sided [-88.20 to -54.87], Standard Error of Mean 8.461
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed model with fixed effects for treatment, visit, treatment-by-visit interaction, baseline value, and a random effect of subject; unstructured covariance matrix was used. Each hypothesis was tested at a significance level of 0.025 (2-sided); Least Square Mean Difference = -52.12, 95% CI 2-sided [-68.70 to -35.55], Standard Error of Mean 8.416

4. Secondary Outcome: Percentage of Participants Achieving at Least a 90% Reduction in PASI (PASI90) at Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percent of BSA affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI90 response was defined as at least a 90% reduction in PASI relative to Baseline.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
percentage of participants | 60.00 (5.903) | 35.23 (5.838) | 3.41 (6.061)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel statistics adjusted for pooled investigator sites was used for the analysis. Each hypothesis was tested at significance level of 0.025 (2-sided); Odds Ratio (OR) = 70.31, 95% CI 2-sided [13.38 to 267.15]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 16.44, 95% CI 2-sided [4.31 to 79.62]

5. Secondary Outcome: Change From Baseline in DLQI Total Score at Week 16
Description: The DLQI is a 10 item general dermatology questionnaire that assesses health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI item response options are rated by the participant from 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life.
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 84 | 84 | 77
scores on a scale | -9.10 (0.635) | -7.03 (0.627) | -1.57 (0.655)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; Week 16. This is a key secondary endpoint; family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant, only then subsequent comparison was tested at the below specified significance level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least square mean difference = -7.52, 95% CI 2-sided [-9.32 to 5.72], Standard Error of Mean 0.913
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least square mean difference = -5.45, 95% CI 2-sided [-7.24 to -3.67], Standard Error of Mean 0.907

6. Secondary Outcome: Percentage of Participants With PGA Score of "Clear" or "Almost Clear" at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
percentage of participants | 37.78 (0.497) | 19.32 (0.493) | 1.14 (0.504)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; This is a key secondary endpoint; family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant,only then subsequent comparison was tested at the below specified significance level; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel statistics adjusted for pooled investigator sites was used for the analysis. Each hypothesis was tested at a significance level of 0.025 (2-sided); Odds Ratio (OR) = 114.40, 95% CI 2-sided [8.95 to 2657.62]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Odds Ratio (OR) = 35.37, 95% CI 2-sided [3.47 to 1084.02]

7. Secondary Outcome: Percentage of Participants Achieving PASI75 Response at Week 4
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least a 75% reduction in PASI relative to Baseline.
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
percentage of participants | 24.44 | 4.55 | 0.00
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; OR and 95% CI not available due to 0% frequency in placebo group
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0386, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; OR and 95% CI not available due to 0% frequency in placebo group

8. Secondary Outcome: Change From Baseline in DLQI Total Score at Week 4
Description: as for outcome 5
Time Frame: Baseline to Week 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 86 | 88 | 83
scores on a scale | -6.03 (0.497) | -5.14 (0.493) | -0.94 (0.504)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; Week 4. This is a key secondary endpoint; family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant, only then subsequent comparison was tested at the below specified significance level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least square mean difference = -5.09, 95% CI 2-sided [-6.49 to -3.70], Standard Error of Mean 0.709
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least square mean difference = -4.20, 95% CI 2-sided [-5.59 to -2.81], Standard Error of Mean 0.706

9. Secondary Outcome: Percent Change From Baseline in Nail Psorasis Severity Index (NAPSI) at Week 16 in Participants With Nail Psoriasis at Baseline
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores represent more severe psoriasis.
Time Frame: Baseline to Week 16
Population: The full analysis population included all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo. Number of participants analyzed signifies those participants who were evaluable (had nail psoriasis at Baseline and had at least one measurement during follow up) for this measure..
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 38 | 38 | 29
percent change | -33.32 (10.518) | -14.98 (10.566) | 7.91 (12.025)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0113, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Least square mean of difference = -41.23, 95% CI 2-sided [-72.91 to -9.54], Standard Error of Mean 15.977
Statistical Analysis 2: Comparison: Tofacitinib 5 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1558, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Least square mean of difference = -22.89, 95% CI 2-sided [-54.64 to 8.86], Standard Error of Mean 16.010

10. Secondary Outcome: Percentage of Participants Maintaining PGA Score of "Clear" or "Almost Clear" at Week 52 Among Participants Achieving PGA Response at Week 16
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). Maintenance of PGA response at Week 52 among patients achieving PGA response at Week 16 is reported. This is a key secondary endpoint. Percentage of participants maintaining the response and the 95% confidence interval (CI) were estimated based on the Kaplan-Meier method. Event is loss of response. Percentage of maintaining response is (1-probability of loss of response).
Time Frame: Week 16 to Week 52
Population: Patients in the full analysis population and those who had PGA response at Week 16 and non-missing post Week 16 data were included. Patients initially treated with placebo were not included as they were advanced to tofacitinib and this maintaining response at Week 52 was not relevant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg
Number analyzed (Participants) | 68 | 46
percentage of participants | 75.00 (0.497) [62.91 to 83.65] | 73.63 (0.493) [58.24 to 84.08]

11. Secondary Outcome: Percentage of Participants Maintaining PASI75 Response at Week 52 Among Participants Achieving PASI75 Response at Week 16
Description: The PASI quantifies severity of a participant's psoriasis based on both lesion severity and percent of BSA affected. PASI is a composite scoring by investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk including axillae and groin, and lower limbs including buttocks), with adjustment for percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response=at least 75% reduction in PASI relative to Baseline. Maintenance of PASI75 response at Week 52 among patients achieving PASI75 response at Week 16 is reported. This is a key secondary endpoint. Probability and the 95% CI were estimated based on the Kaplan-Meier method. Event is loss of response. Percentage of maintaining response is (1-probability of loss of response).
Time Frame: Week 16 to Week 52
Population: Patients in the full analysis population and those who had PASI75 response at Week 16 and non-missing post Week 16 data were included. Patients initially treated with placebo were not included as they were advanced to tofacitinib and this maintaining response at Week 52 was not relevant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg
Number analyzed (Participants) | 73 | 48
percentage of participants | 84.93 (0.497) [74.44 to 91.36] | 76.82 (0.493) [62.04 to 86.44]

12. Secondary Outcome: Percentage of Participants Maintaining PASI90 Response at Week 52 Among Participants Achieving PASI90 at Week 16
Description: The PASI quantifies severity of a participant's psoriasis based on both lesion severity and percent of BSA affected. PASI is a composite scoring by investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk including axillae and groin, and lower limbs including buttocks), with adjustment for percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI90 response=at least 90% reduction in PASI relative to Baseline. Maintenance of PASI90 response at Week 52 among patients achieving PASI90 response at Week 16 is reported. This is a key secondary endpoint. Probability and the 95% CI were estimated based on the Kaplan-Meier method. Event is loss of response. Percentage of maintaining response is (1-probability of loss of response).
Time Frame: Week 16 to Week 52
Population: Patients in the full analysis population and those who had PASI90 response at Week 16 and non-missing post Week 16 data were included. Patients initially treated with placebo were not included as they were advanced to tofacitinib and this maintaining response at Week 52 was not relevant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg
Number analyzed (Participants) | 54 | 31
percentage of participants | 74.07 (0.497) [60.19 to 83.75] | 70.45 (0.493) [50.85 to 83.41]

13. Secondary Outcome: Time to PGA Response up to Week 16
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). Median time to achieve a PGA response up to week 16 is reported. The median time to event was estimated based on the probability of event-rate based on life table estimates (not the observed rate as in outcome measure 1). Median time to event is not estimable if less than 50% of participants had PGA response by Week 16.
Time Frame: Baseline to Week 16
Population: Participants with non-missing post-baseline response data in the full analysis population (all participants who were randomized to the study and received at least 1 dose of study drug) were included.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 88 | 88 | 86
weeks | 8.0 [4.0 to 8.0] | 14.0 [12.0 to NA] — Upper limit of the CI is not estimable. The time frame from Baseline to Week 16 is insufficient to observe the required number of responders for the upper limit. | NA [NA to NA] — Not estimable. Less than half of the participants are responders by Week 16 (ie. censoring percent is >50%).

14. Secondary Outcome: Time to PASI75 Response up to Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least 75% reduction in PASI relative to Baseline. The median time to event was estimated based on the probability of event-rate based on life table estimates (not the observed rate as in outcome measure 2). Median time to event is not estimable if less than 50% of participants had PASI50 response by Week 16.
Time Frame: Baseline up to Week 16
Population: Participants with non-missing post-baseline responses data in the full analysis population (all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo) were included.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 88 | 88 | 86
weeks | 8.0 [8.0 to 12.0] | 16.0 [12.0 to NA] — Upper limit of the CI is not estimable. The time frame from Baseline to Week 16 is insufficient to observe the required number of responders for the upper limit. | NA [NA to NA] — Not estimable. Less than half of the participants are responders by Week 16 (ie. censoring percent is >50%).

15. Secondary Outcome: Time to PASI50 Response up to Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 50 response was defined as at least 50% reduction in PASI relative to Baseline. The median time to event was estimated based on the probability of event-rate based on life table estimates (not the observed rate as in outcome measure 26). Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Baseline up to Week 16
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 88 | 88 | 86
weeks | 4.0 [4.0 to 8.0] | 8.0 [8.0 to 12.0] | NA [NA to NA] — Not estimable. Less than half of the participants are responders by Week 16 (ie. censoring percent is >50%).

16. Secondary Outcome: Percentage of Participants With PGA Response of 'Clear' or 'Almost Clear' Over Time Through Week 52
Description: as for outcome 1
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Week 2 | 3.33 [0.00 to 7.04] | 2.27 [0.00 to 5.39] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 4 | 37.78 [27.76 to 47.79] | 19.32 [11.07 to 27.57] | 2.27 [0.00 to 6.68] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 8 | 57.78 [47.57 to 67.98] | 38.64 [28.46 to 48.81] | 11.36 [1.99 to 20.74] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 12 | 74.44 [65.43 to 83.46] | 50.00 [39.55 to 60.45] | 25.00 [12.21 to 37.79] | 6.82 [0.00 to 14.27]
  Week 16 | 75.56 [66.68 to 84.43] | 52.27 [41.84 to 62.71] | 29.55 [16.06 to 43.03] | 9.09 [0.60 to 17.59]
  Week 20 | 75.56 [66.68 to 84.43] | 54.55 [44.14 to 64.95] | 59.09 [44.56 to 73.62] | 47.73 [32.97 to 62.49]
  Week 32 | 73.33 [64.20 to 82.47] | 53.41 [42.99 to 63.83] | 68.18 [54.42 to 81.94] | 52.27 [37.51 to 67.03]
  Week 40 | 72.22 [62.97 to 81.48] | 55.68 [45.30 to 66.06] | 65.91 [51.90 to 79.92] | 54.55 [39.83 to 69.26]
  Week 52 | 67.78 [58.12 to 77.43] | 54.55 [44.14 to 64.95] | 59.09 [44.56 to 73.62] | 50.00 [35.23 to 64.77]

17. Secondary Outcome: Percentage of Participants in Each PGA Category Over Time Through Week 52
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). Percentage of participants with each PGA score is reported.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: The full analysis population included all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo; n=number of evaluable participants at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Baseline: Clear (n=90,88,44,44) | 0 [95.67 to 100.0] | 0 [83.16 to 99.45] | 0 | 0
  Baseline: Almost Clear (n=90,88,44,44) | 0 | 0 | 0 | 0
  Baseline: Mild (n=90,88,44,44) | 0 | 0 | 0 | 0
  Baseline: Moderate (n=90,88,44,44) | 85.6 | 87.5 | 81.8 | 70.5
  Baseline: Severe (n=90,88,44,44) | 14.4 | 12.5 | 18.2 | 29.5
  Week 2: Clear (n=88,86,44,42) | 0 | 0 | 0 | 0
  Week 2: Almost Clear (n=88,86,44,42) | 3.4 | 2.3 | 0 | 0
  Week 2: Mild (n=88,86,44,42) | 47.7 | 36.0 | 11.4 | 4.8
  Week 2: Moderate (n=88,86,44,42) | 40.9 | 55.8 | 75.0 | 71.4
  Week 2: Severe (n=88,86,44,42) | 8.0 | 5.8 | 13.6 | 23.8
  Week 4: Clear (n=87,88,43,42) | 2.3 | 1.1 | 0 | 0
  Week 4: Almost Clear (n=87,88,43,42) | 36.8 | 18.2 | 2.3 | 0
  Week 4: Mild (n=87,88,43,42) | 29.9 | 39.8 | 23.3 | 14.3
  Week 4: Moderate (n=87,88,43,42) | 27.6 | 36.4 | 53.5 | 69.0
  Week 4: Severe (n=87,88,43,42) | 3.4 | 4.5 | 20.9 | 16.7
  Week 8: Clear (n=85,88,40,39) | 23.5 | 3.4 | 0 | 0
  Week 8: Almost Clear (n=85,88,40,39) | 37.6 | 35.2 | 12.5 | 0
  Week 8: Mild (n=85,88,40,39) | 20.0 | 28.4 | 30.0 | 25.6
  Week 8: Moderate (n=85,88,40,39) | 17.6 | 30.7 | 42.5 | 61.5
  Week 8: Severe (n=85,88,40,39) | 1.2 | 2.3 | 15.0 | 12.8
  Week 12: Clear (n=84,88,40,39) | 34.5 | 12.5 | 0 | 0
  Week 12: Almost Clear (n=84,88,40,39) | 45.2 | 37.5 | 27.5 | 7.7
  Week 12: Mild (n=84,88,40,39) | 11.9 | 27.3 | 30.0 | 30.8
  Week 12: Moderate (n=84,88,40,39) | 6.0 | 22.7 | 37.5 | 51.3
  Week 12: Severe (n=84,88,40,39) | 2.4 | 0 | 5.0 | 10.3
  Week 16: Clear (n=84,84,38,39) | 42.9 | 16.7 | 5.3 | 0
  Week 16: Almost Clear (n=84,84,38,39) | 38.1 | 38.1 | 28.9 | 10.3
  Week 16: Mild (n=84,84,38,39) | 9.5 | 21.4 | 26.3 | 30.8
  Week 16: Moderate (n=84,84,38,39) | 9.5 | 23.8 | 34.2 | 51.3
  Week 16: Severe (n=84,84,38,39) | 0 | 0 | 5.3 | 7.7
  Week 20: Clear (n=84,84,38,39) | 50.0 | 25.0 | 15.8 | 2.6
  Week 20: Almost Clear (n=84,84,38,39) | 31.0 | 32.1 | 52.6 | 51.3
  Week 20: Mild (n=84,84,38,39) | 11.9 | 29.8 | 18.4 | 38.5
  Week 20: Moderate (n=84,84,38,39) | 7.1 | 13.1 | 13.2 | 7.7
  Week 20: Severe (n=84,84,38,39) | 0 | 0 | 0 | 0
  Week 32: Clear (n=83,83,38,37) | 51.8 | 31.3 | 44.7 | 29.7
  Week 32: Almost Clear (n=83,83,38,37) | 27.7 | 25.3 | 34.2 | 32.4
  Week 32: Mild (n=83,83,38,37) | 13.3 | 26.5 | 18.4 | 32.4
  Week 32: Moderate (n=83,83,38,37) | 7.2 | 16.9 | 2.6 | 5.4
  Week 32: Severe (n=83,83,38,37) | 0 | 0 | 0 | 0
  Week 40: Clear (n=81,81,37,36) | 53.1 | 29.6 | 48.6 | 36.1
  Week 40: Almost Clear (n=81,81,37,36) | 27.2 | 30.9 | 29.7 | 30.6
  Week 40: Mild (n=81,81,37,36) | 13.6 | 25.9 | 13.5 | 19.4
  Week 40: Moderate (n=81,81,37,36) | 6.2 | 13.6 | 8.1 | 13.9
  Week 40: Severe (n=81,81,37,36) | 0 | 0 | 0 | 0
  Week 52: Clear (n=80,78,36,36) | 45.0 | 25.6 | 50.0 | 30.6
  Week 52: Almost Clear (n=80,78,36,36) | 31.3 | 35.9 | 22.2 | 30.6
  Week 52: Mild (n=80,78,36,36) | 16.3 | 19.2 | 16.7 | 30.6
  Week 52: Moderate (n=80,78,36,36) | 7.5 | 17.9 | 11.1 | 8.3
  Week 52: Severe (n=80,78,36,36) | 0 | 1.3 | 0 | 0

18. Secondary Outcome: Percentage of Participants Achieving PASI75 Response Over Time Through Week 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least 75% reduction in PASI relative to Baseline. Percentage of participants with PASI 75 response is reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Week 2 | 1.11 [0.00 to 3.28] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 4 | 24.44 [15.57 to 33.32] | 4.55 [0.19 to 8.90] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 8 | 51.11 [40.78 to 61.44] | 31.82 [22.09 to 41.55] | 2.27 [0.00 to 6.68] | 2.27 [0.00 to 6.68]
  Week 12 | 72.22 [62.97 to 81.48] | 47.73 [37.29 to 58.16] | 11.36 [1.99 to 20.74] | 2.27 [0.00 to 6.68]
  Week 16 | 81.11 [73.02 to 89.20] | 54.55 [44.14 to 64.95] | 20.45 [8.54 to 32.37] | 4.55 [0.00 to 10.70]
  Week 20 | 83.33 [75.63 to 91.03] | 54.55 [44.14 to 64.95] | 52.27 [37.51 to 67.03] | 27.27 [14.11 to 40.43]
  Week 32 | 81.11 [73.02 to 89.20] | 59.09 [48.82 to 69.36] | 75.00 [62.21 to 87.79] | 65.91 [51.90 to 79.92]
  Week 40 | 80.00 [71.74 to 88.26] | 56.82 [46.47 to 67.17] | 68.18 [54.42 to 81.94] | 65.91 [51.90 to 79.92]
  Week 52 | 76.67 [67.93 to 85.40] | 59.09 [48.82 to 69.36] | 63.64 [49.42 to 77.85] | 59.09 [44.56 to 73.62]

19. Secondary Outcome: Actual PASI Scores Over Time Through Week 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, 52
Population: The full analysis population included all participants who were randomized to the study and received at least 1 dose of tofacitinib or placebo; number of participants analyzed was the evaluable participants for the specific criteria; n=number of evaluable participants at the specified time point.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Baseline (n=90,88,44,44) | 25.34 (9.106) [0.00 to 3.28] | 25.32 (10.185) [NA to NA] | 25.62 (10.429) [NA to NA] | 26.51 (8.525) [NA to NA]
  Week 2 (n=88,86,44,42) | 19.03 (9.392) [15.57 to 33.32] | 21.23 (9.979) [0.19 to 8.90] | 25.72 (10.582) [NA to NA] | 26.34 (9.456) [NA to NA]
  Week 4 (n=87,88,43,42) | 13.81 (9.826) [40.78 to 61.44] | 17.41 (10.565) [22.09 to 41.55] | 24.81 (12.081) [0.00 to 6.68] | 24.65 (9.433) [0.00 to 6.68]
  Week 8 (n=85,88,40,39) | 8.18 (9.075) [62.97 to 81.48] | 12.56 (10.623) [37.29 to 58.16] | 21.38 (11.689) [1.99 to 20.74] | 22.46 (8.966) [0.00 to 6.68]
  Week 12 (n=84,88,40,39) | 4.56 (6.979) [73.02 to 89.20] | 10.10 (9.858) [44.14 to 64.95] | 17.83 (10.503) [8.54 to 32.37] | 21.35 (9.477) [0.00 to 10.70]
  Week 16 (n=84,84,38,39) | 3.48 (6.722) [75.63 to 91.03] | 8.42 (9.800) [44.14 to 64.95] | 15.27 (11.441) [37.51 to 67.03] | 20.64 (9.738) [14.11 to 40.43]
  Week 20 (84,84,38,39) | 2.75 (5.610) [73.02 to 89.20] | 7.13 (8.280) [48.82 to 69.36] | 6.52 (6.512) [62.21 to 87.79] | 10.43 (7.612) [51.90 to 79.92]
  Week 32 (n=83,83,38,37) | 2.15 (3.810) [71.74 to 88.26] | 6.23 (7.817) [46.47 to 67.17] | 3.09 (5.434) [54.42 to 81.94] | 4.82 (5.517) [51.90 to 79.92]
  Week 40 (n=81,81,37,36) | 2.04 (3.553) [67.93 to 85.40] | 5.74 (6.415) [48.82 to 69.36] | 2.79 (4.458) [49.42 to 77.85] | 3.74 (4.540) [44.56 to 73.62]
  Week 52 (n=80,78,36,36) | 2.82 (4.674) | 6.00 (7.313) | 3.11 (5.027) | 4.69 (4.607)

20. Secondary Outcome: Change From Baseline in PASI Over Time Through Week 52
Description: as for outcome 19
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Week 2 (n=88,86,44,42) | -6.40 (6.724) [15.57 to 33.32] | -4.26 (5.231) [0.19 to 8.90] | 0.10 (4.715) [NA to NA] | -0.04 (3.676) [NA to NA]
  Week 4 (n=87,88,43,42) | -11.74 (8.528) [40.78 to 61.44] | -7.91 (7.053) [22.09 to 41.55] | -0.76 (7.423) [0.00 to 6.68] | -1.72 (3.799) [0.00 to 6.68]
  Week 8 (n=85,88,40,39) | -17.25 (10.244) [62.97 to 81.48] | -12.76 (10.033) [37.29 to 58.16] | -4.25 (8.996) [1.99 to 20.74] | -4.51 (6.130) [0.00 to 6.68]
  Week 12 (n=84,88,40,39) | -20.98 (9.612) [73.02 to 89.20] | -15.22 (11.214) [44.14 to 64.95] | -7.71 (10.717) [8.54 to 32.37] | -5.62 (7.169) [0.00 to 10.70]
  Week 16 (n=84,84,38,39) | -22.07 (10.127) [75.63 to 91.03] | -17.12 (11.711) [44.14 to 64.95] | -10.03 (12.976) [37.51 to 67.03] | -6.33 (8.973) [14.11 to 40.43]
  Week 20 (n=84,84,38,39) | -22.79 (9.675) [73.02 to 89.20] | -18.42 (10.955) [48.82 to 69.36] | -18.79 (12.428) [62.21 to 87.79] | -16.54 (8.732) [51.90 to 79.92]
  Week 32 (n=83,83,38,37) | -23.45 (9.369) [71.74 to 88.26] | -19.45 (10.312) [46.47 to 67.17] | -22.22 (11.550) [54.42 to 81.94] | -21.86 (9.283) [51.90 to 79.92]
  Week 40 (n=81,81,37,36) | -23.47 (9.702) [67.93 to 85.40] | -20.11 (10.292) [48.82 to 69.36] | -22.80 (11.268) [49.42 to 77.85] | -22.94 (9.512) [44.56 to 73.62]
  Week 52 (n=80,78,36,36) | -22.71 (10.655) | -20.04 (10.819) | -22.54 (12.368) | -22.00 (9.429)

21. Secondary Outcome: PASI Component Scores Over Time Through Week 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of BSA" affected. Basic characteristics of psoriatic lesions: erythema, induration, and scaling (PASI components) are scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]) according to a 5-point scale: 0 (no involvement); 1 (slight); 2 (moderate); 3 (marked); 4 (very marked). PASI component score range from 0 to 4, where higher scores indicate greater severity of psoriatic lesions.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Baseline: Erythema (Head/Neck) n=90,88,44,44 | 2.31 (0.830) [15.57 to 33.32] | 2.18 (0.977) [0.19 to 8.90] | 2.18 (1.018) [NA to NA] | 2.39 (0.868) [NA to NA]
  Week 2: Erythema (Head/Neck) n=88,86,44,42 | 1.74 (0.903) [40.78 to 61.44] | 1.77 (1.037) [22.09 to 41.55] | 2.05 (1.033) [0.00 to 6.68] | 2.50 (0.834) [0.00 to 6.68]
  Week 4: Erythema (Head/Neck) n=87,88,43,42 | 1.37 (0.978) [62.97 to 81.48] | 1.44 (1.015) [37.29 to 58.16] | 1.91 (1.065) [1.99 to 20.74] | 2.24 (0.726) [0.00 to 6.68]
  Week 8: Erythema (Head/Neck) n=85,88,40,39 | 0.93 (0.997) [73.02 to 89.20] | 1.14 (1.052) [44.14 to 64.95] | 1.93 (1.141) [8.54 to 32.37] | 2.05 (1.075) [0.00 to 10.70]
  Week 12: Erythema (Head/Neck) n=84,88,40,39 | 0.68 (0.867) [75.63 to 91.03] | 0.94 (1.065) [44.14 to 64.95] | 1.75 (1.171) [37.51 to 67.03] | 1.97 (1.038) [14.11 to 40.43]
  Week 16: Erythema (Head/Neck) n=84,84,38,39 | 0.58 (0.839) [73.02 to 89.20] | 0.82 (1.032) [48.82 to 69.36] | 1.47 (1.156) [62.21 to 87.79] | 1.82 (1.073) [51.90 to 79.92]
  Week 20: Erythema (Head/Neck) n=84,84,38,39 | 0.50 (0.784) [71.74 to 88.26] | 0.82 (0.971) [46.47 to 67.17] | 0.76 (0.883) [54.42 to 81.94] | 1.08 (0.839) [51.90 to 79.92]
  Week 32: Erythema (Head/Neck) n=83,83,38,37 | 0.58 (0.885) [67.93 to 85.40] | 0.73 (0.989) [48.82 to 69.36] | 0.45 (0.860) [49.42 to 77.85] | 0.84 (1.041) [44.56 to 73.62]
  Week 40: Erythema (Head/Neck) n=81,81,37,36 | 0.51 (0.882) | 0.74 (0.946) | 0.43 (0.728) | 0.64 (0.899)
  Week 52: Erythema (Head/Neck) n=80,78,36,36 | 0.58 (0.925) | 0.72 (0.966) | 0.47 (0.774) | 0.78 (0.929)
  Baseline: Erythema (Upper Limbs) n=90,88,44,44 | 2.70 (0.694) | 2.78 (0.686) | 2.66 (0.805) | 2.73 (0.624)
  Week 2: Erythema (Upper Limbs) n=88,86,44,42 | 2.06 (0.793) | 2.28 (0.792) | 2.68 (0.829) | 2.90 (0.692)
  Week 4: Erythema (Upper Limbs) n=87,88,43,42 | 1.61 (0.826) | 1.88 (0.920) | 2.53 (0.960) | 2.71 (0.673)
  Week 8: Erythema (Upper Limbs) n=85,88,40,39 | 1.05 (0.937) | 1.47 (0.982) | 2.35 (1.075) | 2.51 (0.823)
  Week 12: Erythema (Upper Limbs) n=84,88,40,39 | 0.60 (0.778) | 1.17 (1.074) | 2.13 (1.067) | 2.36 (0.873)
  Week 16: Erythema (Upper Limbs) n=84,84,38,39 | 0.51 (0.784) | 0.99 (1.024) | 1.71 (1.137) | 2.33 (0.927)
  Week 20: Erythema (Upper Limbs) n=84,84,38,39 | 0.40 (0.793) | 0.93 (0.967) | 0.97 (0.788) | 1.38 (0.877)
  Week 32: Erythema (Upper Limbs) n=83,83,38,37 | 0.40 (0.697) | 0.96 (1.087) | 0.55 (0.760) | 0.86 (1.004)
  Week 40: Erythema (Upper Limbs) n=81,81,37,36 | 0.44 (0.791) | 0.93 (1.034) | 0.59 (0.927) | 0.78 (0.866)
  Week 52: Erythema (Upper Limbs) n=80,78,36,36 | 0.56 (0.939) | 0.95 (1.031) | 0.69 (0.980) | 0.89 (1.063)
  Baseline: Erythema (Trunk) n=90,88,44,44 | 2.86 (0.696) | 2.81 (0.658) | 2.86 (0.510) | 2.93 (0.625)
  Week 2: Erythema (Trunk) n=88,86,44,42 | 2.28 (0.830) | 2.44 (0.776) | 2.84 (0.568) | 3.05 (0.697)
  Week 4: Erythema (Trunk) n=87,88,43,42 | 1.82 (0.922) | 2.05 (0.883) | 2.72 (0.734) | 2.83 (0.660)
  Week 8: Erythema (Trunk) n=85,88,40,39 | 1.20 (1.056) | 1.65 (1.006) | 2.50 (0.987) | 2.64 (0.778)
  Week 12: Erythema (Trunk) n=84,88,40,39 | 0.81 (1.024) | 1.44 (1.133) | 2.20 (1.137) | 2.54 (0.790)
  Week 16: Erythema (Trunk) n=84,84,38,39 | 0.63 (0.929) | 1.21 (1.173) | 1.87 (1.234) | 2.64 (0.811)
  Week 20: Erythema (Trunk) n=84,84,38,39 | 0.62 (1.005) | 1.12 (1.080) | 1.08 (0.997) | 1.31 (0.800)
  Week 32: Erythema (Trunk) n=83,83,38,37 | 0.58 (0.952) | 1.02 (1.137) | 0.53 (0.893) | 0.70 (0.968)
  Week 40: Erythema (Trunk) n=81,81,37,36 | 0.48 (0.823) | 0.96 (1.078) | 0.43 (0.835) | 0.67 (0.862)
  Week 52: Erythema (Trunk) n=80,78,36,36 | 0.59 (0.924) | 0.99 (1.099) | 0.64 (1.073) | 0.92 (0.937)
  Baseline: Erythema (Lower Limbs) n=90,88,44,44 | 3.03 (0.678) | 2.98 (0.660) | 3.05 (0.746) | 3.16 (0.608)
  Week 2: Erythema (Lower Limbs) n=88,86,44,42 | 2.53 (0.870) | 2.60 (0.830) | 3.05 (0.776) | 3.24 (0.576)
  Week 4: Erythema (Lower Limbs) n=87,88,43,42 | 1.97 (0.946) | 2.23 (0.854) | 2.93 (0.856) | 3.07 (0.677)
  Week 8: Erythema (Lower Limbs) n=85,88,40,39 | 1.33 (1.051) | 1.78 (1.077) | 2.70 (0.939) | 2.92 (0.739)
  Week 12: Erythema (Lower Limbs) n=84,88,40,39 | 0.79 (0.865) | 1.53 (1.082) | 2.48 (1.012) | 2.82 (0.756)
  Week 16: Erythema (Lower Limbs) n=84,84,38,39 | 0.67 (0.883) | 1.44 (1.155) | 2.13 (1.166) | 2.77 (0.810)
  Week 20: Erythema (Lower Limbs) n=84,84,38,39 | 0.54 (0.870) | 1.26 (1.043) | 1.16 (0.945) | 1.77 (0.842)
  Week 32: Erythema (Lower Limbs) n=83,83,38,37 | 0.47 (0.860) | 1.13 (1.197) | 0.66 (0.909) | 1.11 (1.100)
  Week 40: Erythema (Lower Limbs) n=81,81,37,36 | 0.52 (0.963) | 1.14 (1.159) | 0.70 (0.968) | 0.81 (0.889)
  Week 52: Erythema (Lower Limbs) n=80,78,36,36 | 0.70 (1.024) | 1.24 (1.281) | 0.78 (1.198) | 0.94 (1.068)
  Baseline: Induration (Head/Neck) n=90,88,44,44 | 2.23 (0.937) | 1.94 (0.998) | 2.07 (1.065) | 2.20 (0.930)
  Week 2: Induration (Head/Neck) n=88,86,44,42 | 1.63 (0.998) | 1.67 (1.011) | 2.00 (1.100) | 2.19 (0.943)
  Week 4: Induration (Head/Neck) n=87,88,43,42 | 1.16 (1.022) | 1.35 (1.073) | 1.74 (1.071) | 2.10 (0.932)
  Week 8: Induration (Head/Neck) n=85,88,40,39 | 0.84 (1.010) | 1.08 (1.074) | 1.55 (0.959) | 1.92 (1.010)
  Week 12: Induration (Head/Neck) n=84,88,40,39 | 0.63 (0.847) | 0.86 (1.008) | 1.40 (0.900) | 1.72 (0.972)
  Week 16: Induration (Head/Neck) n=84,84,38,39 | 0.51 (0.736) | 0.73 (0.974) | 1.29 (0.984) | 1.56 (0.995)
  Week 20: Induration (Head/Neck) n=84,84,38,39 | 0.40 (0.642) | 0.67 (0.910) | 0.58 (0.683) | 0.90 (0.718)
  Week 32: Induration (Head/Neck) n=83,83,38,37 | 0.49 (0.755) | 0.57 (0.814) | 0.32 (0.702) | 0.62 (0.794)
  Week 40: Induration (Head/Neck) n=81,81,37,36 | 0.44 (0.742) | 0.60 (0.801) | 0.35 (0.633) | 0.53 (0.810)
  Week 52: Induration (Head/Neck) n=80,78,36,36 | 0.53 (0.871) | 0.60 (0.888) | 0.44 (0.735) | 0.61 (0.871)
  Baseline: Induration (Upper Limbs) n=90,88,44,44 | 2.71 (0.738) | 2.59 (0.783) | 2.57 (0.925) | 2.77 (0.677)
  Week 2: Induration (Upper Limbs) n=88,86,44,42 | 2.02 (0.884) | 2.16 (0.919) | 2.52 (0.876) | 2.74 (0.798)
  Week 4: Induration (Upper Limbs) n=87,88,43,42 | 1.54 (1.054) | 1.82 (1.012) | 2.35 (1.021) | 2.62 (0.795)
  Week 8: Induration (Upper Limbs) n=85,88,40,39 | 1.01 (1.029) | 1.40 (1.078) | 2.03 (1.050) | 2.36 (0.903)
  Week 12: Induration (Upper Limbs) n=84,88,40,39 | 0.55 (0.813) | 1.13 (1.081) | 1.78 (1.000) | 2.23 (0.842)
  Week 16: Induration (Upper Limbs) n=84,84,38,39 | 0.39 (0.761) | 1.05 (1.108) | 1.55 (1.083) | 2.08 (0.870)
  Week 20: Induration (Upper Limbs) n=84,84,38,39 | 0.37 (0.818) | 0.90 (1.013) | 0.89 (0.924) | 1.18 (0.823)
  Week 32: Induration (Upper Limbs) n=83,83,38,37 | 0.42 (0.798) | 0.96 (1.064) | 0.58 (0.919) | 0.78 (0.917)
  Week 40: Induration (Upper Limbs) n=81,81,37,36 | 0.47 (0.867) | 0.94 (1.041) | 0.49 (0.768) | 0.75 (0.841)
  Week 52: Induration (Upper Limbs) n=80,78,36,36 | 0.53 (0.886) | 0.90 (0.988) | 0.58 (0.874) | 0.81 (0.951)
  Baseline: Induration (Trunk) n=90,88,44,44 | 2.90 (0.619) | 2.74 (0.703) | 2.91 (0.772) | 2.93 (0.695)
  Week 2: Induration (Trunk) n=88,86,44,42 | 2.25 (0.913) | 2.33 (0.804) | 2.89 (0.689) | 2.90 (0.759)
  Week 4: Induration (Trunk) n=87,88,43,42 | 1.71 (1.109) | 1.95 (0.970) | 2.67 (0.919) | 2.71 (0.742)
  Week 8: Induration (Trunk) n=85,88,40,39 | 1.13 (1.142) | 1.51 (1.061) | 2.25 (1.080) | 2.54 (0.969)
  Week 12: Induration (Trunk) n=84,88,40,39 | 0.73 (1.034) | 1.35 (1.115) | 2.00 (1.109) | 2.33 (0.898)
  Week 16: Induration (Trunk) n=84,84,38,39 | 0.56 (0.961) | 1.15 (1.156) | 1.79 (1.298) | 2.18 (0.942)
  Week 20: Induration (Trunk) n=84,84,38,39 | 0.50 (0.976) | 1.01 (1.070) | 0.97 (0.972) | 1.13 (0.833)
  Week 32: Induration (Trunk) n=83,83,38,37 | 0.49 (0.846) | 0.96 (1.087) | 0.50 (0.980) | 0.70 (0.939)
  Week 40: Induration (Trunk) n=81,81,37,36 | 0.49 (0.910) | 0.89 (1.037) | 0.38 (0.861) | 0.81 (1.091)
  Week 52: Induration (Trunk) n=80,78,36,36 | 0.55 (0.899) | 0.83 (1.012) | 0.50 (0.941) | 0.97 (1.028)
  Baseline: Induration (Lower Limbs) n=90,88,44,44 | 3.03 (0.678) | 2.88 (0.708) | 3.02 (0.821) | 3.16 (0.680)
  Week 2: Induration (Lower Limbs) n=88,86,44,42 | 2.39 (0.915) | 2.43 (0.888) | 2.93 (0.846) | 3.00 (0.826)
  Week 4: Induration (Lower Limbs) n=87,88,43,42 | 1.83 (1.102) | 2.09 (0.978) | 2.81 (0.932) | 2.93 (0.808)
  Week 8: Induration (Lower Limbs) n=85,88,40,39 | 1.22 (1.138) | 1.61 (1.044) | 2.43 (1.035) | 2.67 (0.927)
  Week 12: Induration (Lower Limbs) n=84,88,40,39 | 0.69 (0.878) | 1.36 (1.063) | 2.15 (0.975) | 2.49 (0.970)
  Week 16: Induration (Lower Limbs) n=84,84,38,39 | 0.54 (0.798) | 1.24 (1.115) | 1.95 (1.138) | 2.46 (0.969)
  Week 20: Induration (Lower Limbs) n=84,84,38,39 | 0.44 (0.827) | 1.07 (1.027) | 1.05 (1.012) | 1.41 (0.785)
  Week 32: Induration (Lower Limbs) n=83,83,38,37 | 0.40 (0.826) | 1.01 (1.088) | 0.58 (0.976) | 0.97 (1.013)
  Week 40: Induration (Lower Limbs) n=81,81,37,36 | 0.46 (0.791) | 0.95 (1.011) | 0.68 (1.029) | 0.78 (0.898)
  Week 52: Induration (Lower Limbs) n=80,78,36,36 | 0.61 (0.907) | 1.03 (1.069) | 0.67 (1.069) | 1.03 (1.134)
  Baseline: Scaling (Head/Neck) n=90,88,44,44 | 2.40 (0.946) | 2.01 (1.011) | 2.25 (1.184) | 2.34 (0.987)
  Week 2: Scaling (Head/Neck) n=88,86,44,42 | 1.67 (1.003) | 1.71 (1.004) | 2.11 (1.185) | 2.40 (0.939)
  Week 4: Scaling (Head/Neck) n=87,88,43,42 | 1.24 (1.131) | 1.41 (1.068) | 1.84 (1.214) | 2.24 (0.906)
  Week 8: Scaling (Head/Neck) n=85,88,40,39 | 0.80 (0.986) | 1.02 (1.039) | 1.48 (1.109) | 2.03 (1.013)
  Week 12: Scaling (Head/Neck) n=84,88,40,39 | 0.64 (0.887) | 0.85 (1.012) | 1.38 (1.030) | 1.82 (0.914)
  Week 16: Scaling (Head/Neck) n=84,84,38,39 | 0.57 (0.811) | 0.76 (1.025) | 1.21 (1.018) | 1.72 (0.999)
  Week 20: Scaling (Head/Neck) n=84,84,38,39 | 0.43 (0.664) | 0.67 (0.841) | 0.58 (0.758) | 0.85 (0.812)
  Week 32: Scaling (Head/Neck) n=83,83,38,37 | 0.48 (0.739) | 0.61 (0.809) | 0.29 (0.654) | 0.70 (0.878)
  Week 40: Scaling (Head/Neck) n=81,81,37,36 | 0.51 (0.839) | 0.67 (0.894) | 0.35 (0.716) | 0.67 (0.956)
  Week 52: Scaling (Head/Neck) n=80,78,36,36 | 0.58 (0.897) | 0.63 (0.884) | 0.36 (0.723) | 0.72 (0.914)
  Baseline: Scaling (Upper Limbs) n=90,88,44,44 | 2.72 (0.779) | 2.60 (0.796) | 2.55 (0.848) | 2.82 (0.724)
  Week 2: Scaling (Upper Limbs) n=88,86,44,42 | 2.00 (0.922) | 2.19 (0.952) | 2.43 (0.900) | 2.62 (0.764)
  Week 4: Scaling (Upper Limbs) n=87,88,43,42 | 1.41 (1.106) | 1.77 (1.047) | 2.28 (1.031) | 2.52 (0.804)
  Week 8: Scaling (Upper Limbs) n=85,88,40,39 | 0.89 (0.939) | 1.35 (1.018) | 1.93 (1.118) | 2.28 (0.887)
  Week 12: Scaling (Upper Limbs) n=84,88,40,39 | 0.56 (0.841) | 1.14 (1.106) | 1.60 (1.033) | 2.23 (0.810)
  Week 16: Scaling (Upper Limbs) n=84,84,38,39 | 0.40 (0.793) | 0.99 (1.070) | 1.50 (1.033) | 1.97 (0.903)
  Week 20: Scaling (Upper Limbs) n=84,84,38,39 | 0.39 (0.807) | 0.86 (0.907) | 0.82 (0.834) | 1.21 (0.833)
  Week 32: Scaling (Upper Limbs) n=83,83,38,37 | 0.36 (0.708) | 0.93 (1.010) | 0.42 (0.642) | 0.81 (0.967)
  Week 40: Scaling (Upper Limbs) n=81,81,37,36 | 0.40 (0.801) | 0.96 (1.006) | 0.41 (0.686) | 0.83 (0.910)
  Week 52: Scaling (Upper Limbs) n=80,78,36,36 | 0.48 (0.763) | 0.95 (0.979) | 0.61 (0.871) | 0.92 (1.052)
  Baseline: Scaling (Trunk) n=90,88,44,44 | 2.72 (0.765) | 2.73 (0.784) | 2.77 (0.677) | 2.93 (0.789)
  Week 2: Scaling (Trunk) n=88,86,44,42 | 2.03 (0.928) | 2.27 (0.938) | 2.66 (0.745) | 2.76 (0.759)
  Week 4: Scaling (Trunk) n=87,88,43,42 | 1.52 (1.109) | 1.92 (0.997) | 2.49 (0.883) | 2.57 (0.770)
  Week 8: Scaling (Trunk) n=85,88,40,39 | 0.95 (1.057) | 1.48 (1.039) | 2.10 (1.008) | 2.38 (0.815)
  Week 12: Scaling (Trunk) n=84,88,40,39 | 0.69 (1.006) | 1.27 (1.132) | 1.73 (1.037) | 2.28 (0.857)
  Week 16: Scaling (Trunk) n=84,84,38,39 | 0.52 (0.938) | 1.02 (1.097) | 1.58 (1.106) | 2.10 (0.882)
  Week 20: Scaling (Trunk) n=84,84,38,37 | 0.49 (0.871) | 0.96 (0.987) | 0.82 (0.955) | 1.13 (0.894)
  Week 32: Scaling (Trunk) n=83,83,38,37 | 0.46 (0.754) | 0.92 (0.953) | 0.39 (0.823) | 0.68 (0.852)
  Week 40: Scaling (Trunk) n=81,81,37,36 | 0.49 (0.882) | 0.91 (0.938) | 0.38 (0.861) | 0.78 (0.989)
  Week 52: Scaling (Trunk) n=80,78,36,36 | 0.55 (0.855) | 0.82 (0.818) | 0.53 (0.971) | 0.89 (0.887)
  Baseline: Scaling (Lower Limbs) n=90,88,44,44 | 2.94 (0.709) | 2.92 (0.776) | 2.84 (0.834) | 3.20 (0.765)
  Week 2: Scaling (Lower Limbs) n=88,86,44,42 | 2.24 (1.017) | 2.40 (0.911) | 2.66 (0.888) | 2.98 (0.841)
  Week 4: Scaling (Lower Limbs) n=87,88,43,42 | 1.72 (1.117) | 2.08 (0.997) | 2.49 (0.960) | 2.76 (0.906)
  Week 8: Scaling (Lower Limbs) n=85,88,40,39 | 1.15 (1.129) | 1.52 (1.093) | 2.20 (1.018) | 2.54 (0.884)
  Week 12: Scaling (Lower Limbs) n=84,88,40,39 | 0.67 (0.896) | 1.32 (1.120) | 2.03 (0.920) | 2.51 (0.885)
  Week 16: Scaling (Lower Limbs) n=84,84,38,39 | 0.46 (0.783) | 1.20 (1.106) | 1.82 (1.062) | 2.38 (0.815)
  Week 20: Scaling (Lower Limbs) n=84,84,38,39 | 0.45 (0.870) | 1.14 (1.020) | 0.95 (0.868) | 1.41 (0.751)
  Week 32: Scaling (Lower Limbs) n=83,83,38,37 | 0.37 (0.760) | 1.08 (1.118) | 0.47 (0.797) | 1.03 (1.013)
  Week 40: Scaling (Lower Limbs) n=81,81,37,36 | 0.53 (0.976) | 1.06 (1.041) | 0.51 (0.731) | 0.83 (1.056)
  Week 52: Scaling (Lower Limbs) n=80,78,36,36 | 0.61 (0.921) | 1.08 (1.042) | 0.67 (1.069) | 1.06 (1.120)

22. Secondary Outcome: Change From Baseline in PASI Component Scores Over Time Through Week 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of body surface area (BSA)" affected. Basic characteristics of psoriatic lesions: erythema, induration, and scaling (PASI components) are scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]) according to a 5-point scale: 0 (no involvement); 1 (slight); 2 (moderate); 3 (marked); 4 (very marked). PASI component score range from 0 to 4, where higher scores indicate greater severity of psoriatic lesions.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Week 2: Erythema (Head/Neck) n=88,86,44,42) | -0.56 (0.676) [40.78 to 61.44] | -0.41 (0.757) [22.09 to 41.55] | -0.14 (0.594) [0.00 to 6.68] | 0.10 (0.532) [0.00 to 6.68]
  Week 4: Erythema (Head/Neck) n=87,88,43,42) | -0.94 (0.854) [62.97 to 81.48] | -0.74 (0.890) [37.29 to 58.16] | -0.26 (0.727) [1.99 to 20.74] | -0.17 (0.621) [0.00 to 6.68]
  Week 8: Erythema (Head/Neck) n=85,88,40,39 | -1.36 (0.962) [73.02 to 89.20] | -1.05 (1.038) [44.14 to 64.95] | -0.20 (1.114) [8.54 to 32.37] | -0.38 (0.935) [0.00 to 10.70]
  Week 12: Erythema (Head/Neck) n=84,88,40,39 | -1.61 (0.957) [75.63 to 91.03] | -1.24 (1.135) [44.14 to 64.95] | -0.38 (1.295) [37.51 to 67.03] | -0.46 (0.942) [14.11 to 40.43]
  Week 16: Erythema (Head/Neck) n=84,84,38,39 | -1.70 (1.015) [73.02 to 89.20] | -1.43 (1.175) [48.82 to 69.36] | -0.66 (1.361) [62.21 to 87.79] | -0.62 (0.907) [51.90 to 79.92]
  Week 20: Erythema (Head/Neck) n=84,84,38,39 | -1.79 (0.945) [71.74 to 88.26] | -1.43 (1.185) [46.47 to 67.17] | -1.37 (1.172) [54.42 to 81.94] | -1.36 (1.158) [51.90 to 79.92]
  Week 32: Erythema (Head/Neck) n=83,83,38,37 | -1.71 (1.030) [67.93 to 85.40] | -1.51 (1.203) [48.82 to 69.36] | -1.68 (1.254) [49.42 to 77.85] | -1.59 (1.257) [44.56 to 73.62]
  Week 40: Erythema (Head/Neck) n=81,81,37,36 | -1.78 (1.084) | -1.51 (1.195) | -1.68 (1.132) | -1.81 (1.191)
  Week 52: Erythema (Head/Neck) n=80,78,36,36 | -1.73 (1.079) | -1.53 (1.181) | -1.61 (1.225) | -1.67 (1.265)
  Week 2: Erythema (Upper Limbs) n=88,86,44,42 | -0.64 (0.698) | -0.51 (0.609) | 0.02 (0.403) | 0.14 (0.417)
  Week 4: Erythema (Upper Limbs) n=87,88,43,42 | -1.09 (0.858) | -0.91 (0.839) | -0.12 (0.697) | -0.05 (0.582)
  Week 8: Erythema (Upper Limbs) n=85,88,40,39 | -1.65 (0.984) | -1.32 (0.977) | -0.28 (0.784) | -0.26 (0.677)
  Week 12: Erythema (Upper Limbs) n=84,88,40,39 | -2.08 (0.908) | -1.61 (1.159) | -0.50 (0.877) | -0.41 (0.818)
  Week 16: Erythema (Upper Limbs) n=84,84,38,39 | -2.17 (1.004) | -1.81 (1.092) | -0.92 (0.941) | -0.44 (0.852)
  Week 20: Erythema (Upper Limbs) n=84,84,38,39 | -2.27 (1.057) | -1.87 (1.117) | -1.66 (0.966) | -1.38 (1.042)
  Week 32: Erythema (Upper Limbs) n=83,83,38,37 | -2.29 (0.957) | -1.83 (1.257) | -2.08 (1.148) | -1.89 (0.994)
  Week 40: Erythema (Upper Limbs) n=81,81,37,36 | -2.26 (1.081) | -1.89 (1.151) | -2.05 (1.153) | -1.94 (1.094)
  Week 52: Erythema (Upper Limbs) n=80,78,36,36 | -2.14 (1.111) | -1.85 (1.185) | -1.94 (1.286) | -1.83 (1.183)
  Week 2: Erythema (Trunk) n=88,86,44,42 | -0.57 (0.724) | -0.41 (0.639) | -0.02 (0.457) | 0.10 (0.370)
  Week 4: Erythema (Trunk) n=87,88,43,42 | -1.05 (0.888) | -0.76 (0.844) | -0.14 (0.774) | -0.12 (0.550)
  Week 8: Erythema (Trunk) n=85,88,40,39 | -1.66 (1.041) | -1.16 (0.969) | -0.35 (0.949) | -0.28 (0.560)
  Week 12: Erythema (Trunk) n=84,88,40,39 | -2.04 (1.092) | -1.36 (1.176) | -0.65 (1.167) | -0.38 (0.711)
  Week 16: Erythema (Trunk) n=84,84,38,39 | -2.21 (1.054) | -1.61 (1.203) | -0.97 (1.262) | -0.28 (0.793)
  Week 20: Erythema (Trunk) n=84,84,38,39 | -2.23 (1.134) | -1.70 (1.200) | -1.76 (1.025) | -1.62 (1.091)
  Week 32: Erythema (Trunk) n=83,83,38,37 | -2.25 (1.034) | -1.80 (1.276) | -2.32 (1.016) | -2.22 (1.004)
  Week 40: Erythema (Trunk) n=81,81,37,36 | -2.36 (1.028) | -1.86 (1.212) | -2.43 (0.929) | -2.22 (1.072)
  Week 52: Erythema (Trunk) n=80,78,36,36 | -2.24 (1.082) | -1.82 (1.256) | -2.22 (1.174) | -1.97 (1.158)
  Week 2: Erythema (Lower Limbs) n=88,86,44,42 | -0.50 (0.587) | -0.38 (0.722) | 0.00 (0.374) | 0.05 (0.379)
  Week 4: Erythema (Lower Limbs) n=87,88,43,42 | -1.07 (0.860) | -0.75 (0.820) | -0.12 (0.625) | -0.12 (0.593)
  Week 8: Erythema (Lower Limbs) n=85,88,40,39 | -1.71 (1.010) | -1.19 (1.123) | -0.33 (0.764) | -0.26 (0.637)
  Week 12: Erythema (Lower Limbs) n=84,88,40,39 | -2.24 (0.965) | -1.44 (1.183) | -0.58 (0.958) | -0.36 (0.778)
  Week 16: Erythema (Lower Limbs) n=84,84,38,39 | -2.36 (1.014) | -1.55 (1.255) | -0.89 (1.085) | -0.41 (0.818)
  Week 20: Erythema (Lower Limbs) n=84,84,38,39 | -2.49 (1.000) | -1.73 (1.274) | -1.87 (0.991) | -1.41 (0.993)
  Week 32: Erythema (Lower Limbs) n=83,83,38,37 | -2.54 (1.028) | -1.86 (1.372) | -2.37 (1.025) | -2.05 (1.129)
  Week 40: Erythema (Lower Limbs) n=81,81,37,36 | -2.52 (1.062) | -1.86 (1.243) | -2.32 (1.082) | -2.33 (1.121)
  Week 52: Erythema (Lower Limbs) n=80,78,36,36 | -2.33 (1.077) | -1.74 (1.400) | -2.25 (1.251) | -2.19 (1.215)
  Week 2: Induration (Head/Neck) n=88,86,44,42 | -0.59 (0.705) | -0.27 (0.602) | -0.07 (0.398) | -0.02 (0.468)
  Week 4: Induration (Head/Neck) n=87,88,43,42 | -1.07 (0.974) | -0.59 (0.892) | -0.30 (0.708) | -0.12 (0.670)
  Week 8: Induration (Head/Neck) n=85,88,40,39 | -1.38 (1.080) | -0.86 (0.937) | -0.50 (1.086) | -0.33 (0.927)
  Week 12: Induration (Head/Neck) n=84,88,40,39 | -1.58 (1.032) | -1.08 (1.031) | -0.65 (1.075) | -0.54 (0.913)
  Week 16: Induration (Head/Neck) n=84,84,38,39 | -1.70 (1.106) | -1.24 (1.060) | -0.76 (1.240) | -0.69 (0.863)
  Week 20: Induration (Head/Neck) n=84,84,38,39 | -1.81 (1.058) | -1.30 (1.084) | -1.47 (1.133) | -1.36 (0.903)
  Week 32: Induration (Head/Neck) n=83,83,38,37 | -1.71 (1.121) | -1.41 (1.094) | -1.74 (1.155) | -1.65 (1.160)
  Week 40: Induration (Head/Neck) n=81,81,37,36 | -1.75 (1.124) | -1.37 (1.066) | -1.68 (1.056) | -1.78 (1.198)
  Week 52: Induration (Head/Neck) n=80,78,36,36 | -1.68 (1.178) | -1.36 (1.139) | -1.58 (1.228) | -1.69 (1.215)
  Week 2: Induration (Upper Limbs) n=88,86,44,42 | -0.68 (0.766) | -0.42 (0.727) | -0.05 (0.526) | -0.07 (0.407)
  Week 4: Induration (Upper Limbs) n=87,88,43,42 | -1.17 (1.048) | -0.77 (0.867) | -0.21 (0.833) | -0.19 (0.707)
  Week 8: Induration (Upper Limbs) n=85,88,40,39 | -1.69 (1.024) | -1.19 (1.092) | -0.55 (1.011) | -0.41 (0.751)
  Week 12: Induration (Upper Limbs) n=84,88,40,39 | -2.17 (0.862) | -1.47 (1.231) | -0.80 (1.091) | -0.54 (0.822)
  Week 16: Induration (Upper Limbs) n=84,84,38,39 | -2.32 (0.867) | -1.52 (1.217) | -1.05 (1.293) | -0.69 (0.977)
  Week 20: Induration (Upper Limbs) n=84,84,38,39 | -2.35 (1.012) | -1.67 (1.186) | -1.71 (1.250) | -1.59 (1.093)
  Week 32: Induration (Upper Limbs) n=83,83,38,37 | -2.29 (1.018) | -1.61 (1.296) | -2.03 (1.150) | -1.97 (1.093)
  Week 40: Induration (Upper Limbs) n=81,81,37,36 | -2.25 (1.067) | -1.65 (1.266) | -2.11 (1.100) | -1.97 (1.108)
  Week 52: Induration (Upper Limbs) n=80,78,36,36 | -2.20 (1.107) | -1.69 (1.282) | -2.03 (1.183) | -1.92 (1.204)
  Week 2: Induration (Trunk) n=88,86,44,42 | -0.65 (0.728) | -0.43 (0.660) | -0.02 (0.457) | -0.05 (0.439)
  Week 4: Induration (Trunk) n=87,88,43,42 | -1.20 (1.044) | -0.78 (0.850) | -0.23 (0.812) | -0.24 (0.576)
  Week 8: Induration (Trunk) n=85,88,40,39 | -1.78 (1.084) | -1.23 (1.003) | -0.68 (1.071) | -0.38 (0.673)
  Week 12: Induration (Trunk) n=84,88,40,39 | -2.19 (1.035) | -1.39 (1.129) | -0.90 (1.194) | -0.59 (0.637)
  Week 16: Induration (Trunk) n=84,84,38,39 | -2.36 (0.965) | -1.57 (1.154) | -1.13 (1.398) | -0.74 (0.785)
  Week 20: Induration (Trunk) n=84,84,38,39 | -2.42 (0.984) | -1.71 (1.071) | -1.95 (1.138) | -1.79 (1.031)
  Week 32: Induration (Trunk) n=83,83,38,37 | -2.41 (0.938) | -1.76 (1.122) | -2.42 (1.222) | -2.22 (1.158)
  Week 40: Induration (Trunk) n=81,81,37,36 | -2.41 (1.058) | -1.84 (1.145) | -2.57 (1.068) | -2.08 (1.360)
  Week 52: Induration (Trunk) n=80,78,36,36 | -2.36 (1.070) | -1.90 (1.180) | -2.47 (1.207) | -1.92 (1.339)
  Week 2: Induration (Lower Limbs) n=88,86,44,42 | -0.65 (0.803) | -0.43 (0.660) | -0.09 (0.421) | -0.14 (0.417)
  Week 4: Induration (Lower Limbs) n=87,88,43,42 | -1.22 (0.993) | -0.78 (0.809) | -0.21 (0.773) | -0.21 (0.415)
  Week 8: Induration (Lower Limbs) n=85,88,40,39 | -1.82 (1.002) | -1.26 (0.977) | -0.60 (0.955) | -0.49 (0.683)
  Week 12: Induration (Lower Limbs) n=84,88,40,39 | -2.36 (0.845) | -1.51 (1.093) | -0.85 (0.975) | -0.67 (0.772)
  Week 16: Induration (Lower Limbs) n=84,84,38,39 | -2.51 (0.814) | -1.63 (1.159) | -1.08 (1.148) | -0.69 (0.766)
  Week 20: Induration (Lower Limbs) n=84,84,38,39 | -2.61 (0.865) | -1.80 (1.039) | -1.97 (1.026) | -1.74 (0.818)
  Week 32: Induration (Lower Limbs) n=83,83,38,37 | -2.64 (0.957) | -1.86 (1.106) | -2.45 (1.083) | -2.14 (1.058)
  Week 40: Induration (Lower Limbs) n=81,81,37,36 | -2.57 (0.974) | -1.93 (1.022) | -2.35 (1.033) | -2.31 (1.064)
  Week 52: Induration (Lower Limbs) n=80,78,36,36 | -2.43 (1.041) | -1.85 (1.140) | -2.39 (1.178) | -2.06 (1.194)
  Week 2: Scaling (Head/Neck) n=88,86,44,42 | -0.72 (0.802) | -0.28 (0.587) | -0.14 (0.594) | 0.05 (0.379)
  Week 4: Scaling (Head/Neck) n=87,88,43,42 | -1.16 (1.077) | -0.60 (0.766) | -0.40 (0.955) | -0.12 (0.633)
  Week 8: Scaling (Head/Neck) n=85,88,40,39 | -1.60 (1.157) | -0.99 (1.000) | -0.75 (1.296) | -0.38 (0.963)
  Week 12: Scaling (Head/Neck) n=84,88,40,39 | -1.76 (1.137) | -1.16 (1.103) | -0.83 (1.338) | -0.59 (0.993)
  Week 16: Scaling (Head/Neck) n=84,84,38,39 | -1.83 (1.160) | -1.31 (1.151) | -0.97 (1.404) | -0.69 (0.977)
  Week 20: Scaling (Head/Neck) n=84,84,38,39 | -1.98 (1.075) | -1.40 (1.110) | -1.61 (1.366) | -1.56 (1.021)
  Week 32: Scaling (Head/Neck) n=83,83,38,37 | -1.92 (1.073) | -1.47 (1.162) | -1.89 (1.290) | -1.70 (1.266)
  Week 40: Scaling (Head/Neck) n=81,81,37,36 | -1.88 (1.198) | -1.41 (1.138) | -1.78 (1.250) | -1.78 (1.267)
  Week 52: Scaling (Head/Neck) n=80,78,36,36 | -1.81 (1.192) | -1.45 (1.202) | -1.78 (1.456) | -1.72 (1.233)
  Week 2: Scaling (Upper Limbs) n=88,86,44,42 | -0.72 (0.843) | -0.41 (0.602) | -0.11 (0.579) | -0.19 (0.634)
  Week 4: Scaling (Upper Limbs) n=87,88,43,42 | -1.31 (1.154) | -0.83 (0.847) | -0.26 (0.848) | -0.29 (0.742)
  Week 8: Scaling (Upper Limbs) n=85,88,40,39 | -1.84 (1.078) | -1.25 (0.950) | -0.63 (1.030) | -0.56 (0.940)
  Week 12: Scaling (Upper Limbs) n=84,88,40,39 | -2.18 (0.894) | -1.47 (1.114) | -0.93 (1.023) | -0.62 (1.016)
  Week 16: Scaling (Upper Limbs) n=84,84,38,39 | -2.33 (0.998) | -1.62 (1.040) | -1.00 (1.115) | -0.87 (1.105)
  Week 20: Scaling (Upper Limbs) n=84,84,38,39 | -2.35 (1.047) | -1.75 (1.005) | -1.68 (1.093) | -1.64 (1.112)
  Week 32: Scaling (Upper Limbs) n=83,83,38,37 | -2.37 (1.009) | -1.67 (1.025) | -2.08 (0.997) | -2.03 (1.258)
  Week 40: Scaling (Upper Limbs) n=81,81,37,36 | -2.32 (1.127) | -1.65 (1.153) | -2.08 (1.064) | -2.00 (1.195)
  Week 52: Scaling (Upper Limbs) n=80,78,36,36 | -2.25 (1.175) | -1.68 (1.201) | -1.89 (1.282) | -1.92 (1.381)
  Week 2: Scaling (Trunk) n=88,86,44,42 | -0.68 (0.810) | -0.49 (0.682) | -0.11 (0.655) | -0.17 (0.490)
  Week 4: Scaling (Trunk) n=87,88,43,42 | -1.22 (1.104) | -0.81 (0.842) | -0.28 (0.934) | -0.36 (0.692)
  Week 8: Scaling (Trunk) n=85,88,40,39 | -1.79 (1.124) | -1.25 (0.997) | -0.70 (1.018) | -0.54 (0.790)
  Week 12: Scaling (Trunk) n=84,88,40,39 | -2.06 (1.045) | -1.45 (1.174) | -1.05 (1.154) | -0.64 (0.932)
  Week 16: Scaling (Trunk) n=84,84,38,39 | -2.23 (1.090) | -1.71 (1.136) | -1.21 (1.255) | -0.82 (0.970)
  Week 20: Scaling (Trunk) n=84,84,38,39 | -2.26 (1.088) | -1.77 (1.090) | -1.97 (1.219) | -1.79 (1.174)
  Week 32: Scaling (Trunk) n=83,83,38,37 | -2.28 (0.992) | -1.82 (1.049) | -2.39 (1.054) | -2.22 (1.250)
  Week 40: Scaling (Trunk) n=81,81,37,36 | -2.22 (1.173) | -1.83 (1.160) | -2.43 (1.042) | -2.11 (1.410)
  Week 52: Scaling (Trunk) n=80,78,36,36 | -2.18 (1.188) | -1.94 (1.049) | -2.31 (1.215) | -2.00 (1.352)
  Week 2: Scaling (Lower Limbs) n=88,86,44,42 | -0.70 (0.846) | -0.51 (0.778) | -0.18 (0.657) | -0.21 (0.565)
  Week 4: Scaling (Lower Limbs) n=87,88,43,42 | -1.22 (1.016) | -0.84 (0.933) | -0.35 (0.997) | -0.43 (0.668)
  Week 8: Scaling (Lower Limbs) n=85,88,40,39 | -1.80 (1.044) | -1.40 (1.078) | -0.63 (1.125) | -0.69 (0.863)
  Week 12: Scaling (Lower Limbs) n=84,88,40,39 | -2.30 (0.915) | -1.60 (1.160) | -0.75 (1.080) | -0.72 (0.916)
  Week 16: Scaling (Lower Limbs) n=84,84,38,39 | -2.50 (0.912) | -1.74 (1.173) | -0.95 (1.293) | -0.85 (1.014)
  Week 20: Scaling (Lower Limbs) n=84,84,38,39 | -2.51 (0.963) | -1.80 (1.138) | -1.82 (1.136) | -1.82 (1.023)
  Week 32: Scaling (Lower Limbs) n=83,83,38,37 | -2.58 (0.964) | -1.86 (1.128) | -2.29 (1.160) | -2.16 (1.236)
  Week 40: Scaling (Lower Limbs) n=81,81,37,36 | -2.40 (1.190) | -1.89 (1.118) | -2.22 (1.004) | -2.33 (1.331)
  Week 52: Scaling (Lower Limbs) n=80,78,36,36 | -2.33 (1.111) | -1.88 (1.151) | -2.08 (1.360) | -2.11 (1.326)

23. Secondary Outcome: Percent Change From Baseline in PASI Scores Over Time Through Week 52
Description: as for outcome 19
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percent change
  Week 2 (n=88,86,44,42) | -24.93 (2.399) [15.57 to 33.32] | -16.28 (2.409) [0.19 to 8.90] | 1.37 (3.392) [NA to NA] | -0.35 (3.473) [NA to NA]
  Week 4 (n=87,88,43,42) | -46.24 (3.135) | -32.47 (3.127) | -1.98 (4.444) | -7.31 (4.527)
  Week 8 (n=85,88,40,39) | -66.96 (3.769) | -51.24 (3.739) | -13.17 (5.384) | -16.18 (5.488)
  Week 12 (n=84,88,40,39) | -80.64 (3.631) | -59.73 (3.585) | -25.13 (5.205) | -20.40 (5.304)
  Week 16 (n=84,84,38,39) | -84.35 (3.912) | -66.69 (3.874) | -32.79 (5.651) | -21.63 (5.721)
  Week 20 (n=84,84,38,39) | -87.89 (3.024) | -71.93 (3.002) | -69.85 (4.399) | -60.85 (4.423)
  Week 32 (n=83,83,38,37) | -90.47 (2.444) | -76.06 (2.437) | -86.63 (3.584) | -81.43 (3.622)
  Week 40 (n=81,81,37,36) | -90.18 (2.264) | -77.29 (2.258) | -87.73 (3.332) | -83.64 (3.368)
  Week 52 (n=80,78,36,36) | -86.05 (2.763) | -75.55 (2.764) | -84.65 (4.066) | -79.27 (4.101)

24. Secondary Outcome: Actual BSA Over Time Through Week 52
Description: as for outcome 3
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent BSA
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percent BSA
  Baseline (n=90,88,44,44) | 36.36 (18.035) [15.57 to 33.32] | 37.41 (19.614) [0.19 to 8.90] | 35.29 (18.294) [NA to NA] | 36.25 (16.018) [NA to NA]
  Week 2 (n=88,86,44,44) | 33.95 (17.537) | 36.56 (19.363) | 36.84 (18.808) | 36.38 (16.592)
  Week 4 (n=87,88,43,42) | 27.82 (18.599) | 32.75 (18.314) | 38.32 (19.355) | 36.30 (16.916)
  Week 8 (n=85,88,40,39) | 17.62 (18.411) | 24.38 (19.583) | 36.75 (19.817) | 34.99 (16.182)
  Week 12 (n=84,88,40,39) | 10.59 (15.486) | 20.45 (20.462) | 33.15 (20.483) | 34.06 (17.142)
  Week 16 (n=84,84,38,39) | 7.57 (13.395) | 16.52 (18.899) | 28.57 (21.645) | 34.54 (18.293)
  Week 20 (n=84,84,38,39) | 5.05 (10.041) | 13.69 (16.976) | 15.50 (16.522) | 24.83 (19.044)
  Week 32 (n=83,83,38,37) | 3.22 (5.894) | 11.47 (16.304) | 6.95 (10.262) | 9.03 (11.781)
  Week 40 (n=81,81,37,36) | 2.56 (5.412) | 10.32 (13.077) | 5.88 (8.351) | 6.35 (9.462)
  Week 52 (n=80,78,36,36) | 3.83 (7.908) | 10.94 (15.255) | 5.00 (7.686) | 7.87 (9.584)

25. Secondary Outcome: Percent Change From Baseline in BSA Over Time Through Week 52
Description: as for outcome 3
Time Frame: Baseline and weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percent change
  Week 2 (n=88,86,44,44) | -5.58 (2.083) | -2.53 (2.093) | 4.79 (2.947) | 2.14 (3.016)
  Week 4 (n=87,88,43,42) | -21.90 (3.202) | -10.98 (3.193) | 10.29 (4.541) | 2.28 (4.622)
  Week 8 (n=85,88,40,39) | -46.98 (4.909) | -33.22 (4.870) | 8.73 (7.017) | -0.42 (7.155)
  Week 12 (n=84,88,40,39) | -65.97 (5.536) | -44.44 (5.471) | 0.41 (7.928) | 0.48 (8.086)
  Week 16 (n=84,84,38,39) | -73.80 (5.903) | -54.41 (5.839) | -8.85 (8.511) | 4.13 (8.632)
  Week 20 (n=84,84,38,39) | -82.65 (4.459) | -62.35 (4.419) | -49.35 (6.495) | -28.86 (6.530)
  Week 32 (n=83,83,38,37) | -87.55 (3.531) | -70.55 (3.521) | -74.83 (5.186) | -73.95 (5.235)
  Week 40 (n=81,81,37,36) | -90.00 (3.213) | -73.00 (3.207) | -79.48 (4.743) | -79.91 (4.786)
  Week 52 (n=80,78,36,36) | -84.16 (3.867) | -72.28 (3.868) | -81.70 (5.681) | -74.02 (5.737)

26. Secondary Outcome: Percentage of Participants With PASI50 Response Over Time Through Week 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 50 response was defined as at least 50% reduction in PASI relative to Baseline. Percentage of participants with PASI50 response is reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Week 2 | 21.11 [12.68 to 29.54] | 5.68 [0.85 to 10.52] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 4 | 48.89 [38.56 to 59.22] | 27.27 [17.97 to 36.58] | 4.55 [0.00 to 10.70] | 4.55 [0.00 to 10.70]
  Week 8 | 74.44 [65.43 to 83.46] | 55.68 [45.30 to 66.06] | 13.64 [3.50 to 23.78] | 4.55 [0.00 to 10.70]
  Week 12 | 81.11 [73.02 to 89.20] | 64.77 [54.79 to 74.75] | 27.27 [14.11 to 40.43] | 9.09 [0.60 to 17.59]
  Week 16 | 86.67 [79.64 to 93.69] | 71.59 [62.17 to 81.01] | 40.91 [26.38 to 55.44] | 18.18 [6.79 to 29.58]
  Week 20 | 85.56 [78.29 to 92.82] | 72.73 [63.42 to 82.03] | 68.18 [54.42 to 81.94] | 63.64 [49.42 to 77.85]
  Week 32 | 88.89 [82.40 to 95.38] | 78.41 [69.81 to 87.01] | 79.55 [67.63 to 91.46] | 75.00 [62.21 to 87.79]
  Week 40 | 87.78 [81.01 to 94.54] | 80.68 [72.43 to 88.93] | 79.55 [67.63 to 91.46] | 72.73 [59.57 to 85.89]
  Week 52 | 83.33 [75.63 to 91.03] | 73.86 [64.68 to 83.04] | 77.27 [64.89 to 89.66] | 75.00 [62.21 to 87.79]

27. Secondary Outcome: Percentage of Participants With PASI90 Response Over Time Through Week 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 90 response was defined as at least 90% reduction in PASI relative to Baseline. Percentage of participants with PASI90 response up to Week 52 is reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Week 2 | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 4 | 7.78 [2.24 to 13.31] | 2.27 [0.00 to 5.39] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 8 | 27.78 [18.52 to 37.03] | 13.64 [6.47 to 20.81] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 12 | 51.11 [40.78 to 61.44] | 29.55 [20.01 to 39.08] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 16 | 60.00 [49.88 to 70.12] | 35.23 [25.25 to 45.21] | 6.82 [0.00 to 14.27] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 20 | 71.11 [61.75 to 80.48] | 35.23 [25.25 to 45.21] | 25.00 [12.21 to 37.79] | 9.09 [0.60 to 17.59]
  Week 32 | 65.56 [55.74 to 75.37] | 42.05 [31.73 to 52.36] | 56.82 [42.18 to 71.45] | 40.91 [26.38 to 55.44]
  Week 40 | 66.67 [56.93 to 76.41] | 35.23 [25.25 to 45.21] | 56.82 [42.18 to 71.45] | 45.45 [30.74 to 60.17]
  Week 52 | 56.67 [46.43 to 66.90] | 38.64 [28.46 to 48.81] | 56.82 [42.18 to 71.45] | 36.36 [22.15 to 50.58]

28. Secondary Outcome: Percentage of Participants With PASI125 Over Time Through Week 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. Percentage of participants with PASI score of at least 125% of baseline PASI score are reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Week 2 (n=88,86,44,42) | 2.27 [0.00 to 5.39] | 1.16 [0.00 to 3.43] | 4.55 [0.00 to 10.70] | 4.76 [0.00 to 11.20]
  Week 4 (n=87,88,43,42) | 2.30 [0.00 to 5.45] | 1.14 [0.00 to 3.35] | 13.95 [3.60 to 24.31] | 2.38 [0.00 to 6.99]
  Week 8 (n=85,88,40,39) | 2.35 [0.00 to 5.58] | 1.14 [0.00 to 3.35] | 17.50 [5.72 to 29.28] | 2.56 [0.00 to 7.52]
  Week 12 (n=84,88,40,39) | 1.19 [0.00 to 3.51] | 1.14 [0.00 to 3.35] | 7.50 [0.00 to 15.66] | 5.13 [0.00 to 12.05]
  Week 16 (n=84,84,38,39) | 1.19 [0.00 to 3.51] | 2.38 [0.00 to 5.64] | 10.53 [0.77 to 20.28] | 7.69 [0.00 to 16.06]
  Week 20 (n=84,84,38,39) | 1.19 [0.00 to 3.51] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 2.56 [0.00 to 7.52]
  Week 32 (n=83,83,38,37) | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 40 (n=81,81,37,36) | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 52 (n=80,78,36,36) | 1.25 [0.00 to 3.68] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.

29. Secondary Outcome: Actual Nail Psoriasis Severity Index (NAPSI) Score Over Time Through Week 52 in Participants With Nail Psoriasis at Baseline
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores represents more severe psoriasis.
Time Frame: Baseline and Weeks 8, 16, 20, 32, 40, and 52
Population: Number of participants analyzed signifies the FAS participants (randomized and received at least 1 dose of investigational drug) who were evaluable (had nail psoriasis at Baseline and at least 1 measurement during follow up) for this measure. n=number of evaluable participants at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 40 | 38 | 18 | 18
units on a scale
  Baseline (n=40,38,18,18) | 25.8 (20.58) [0.00 to 5.58] | 26.2 (16.97) [0.00 to 3.35] | 28.7 (21.90) [5.72 to 29.28] | 25.2 (16.37) [0.00 to 7.52]
  Week 8 (n=39,38,15,15) | 23.0 (19.45) [0.00 to 3.51] | 23.6 (17.29) [0.00 to 5.64] | 28.6 (23.66) [0.77 to 20.28] | 30.7 (18.48) [0.00 to 16.06]
  Week 16 (n=38,38,14,15) | 17.2 (19.14) [0.00 to 3.51] | 19.8 (18.30) [NA to NA] | 30.3 (23.86) [NA to NA] | 28.9 (20.54) [0.00 to 7.52]
  Week 20 (n=37,38,14,15) | 13.9 (18.70) [NA to NA] | 17.2 (16.94) [NA to NA] | 28.6 (24.02) [NA to NA] | 30.1 (19.08) [NA to NA]
  Week 32 (n=37,37,14,14) | 12.6 (19.59) [NA to NA] | 15.5 (16.69) [NA to NA] | 16.2 (18.48) [NA to NA] | 17.1 (12.69) [NA to NA]
  Week 40 (n=36,36,13,13) | 9.6 (18.65) [0.00 to 3.68] | 14.9 (16.01) [NA to NA] | 15.7 (15.82) [NA to NA] | 14.5 (13.93) [NA to NA]
  Week 52 (n=31,34,12,13) | 10.0 (20.22) | 13.2 (17.96) | 13.8 (18.54) | 10.5 (12.67)

30. Secondary Outcome: Change From Baseline in NAPSI Over Time Through Week 52 in Participants With Nail Psoriasis at Baseline
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail was divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores represents more severe psoriasis.
Time Frame: Baseline and weeks 8, 16, 20, 32, 40, and 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 40 | 38 | 18 | 18
units on a scale
  Week 8 (n=39,38,15,15) | -3.60 (1.416) [0.00 to 3.51] | -2.76 (1.434) [0.00 to 5.64] | 2.17 (2.282) [0.77 to 20.28] | 2.64 (2.283) [0.00 to 16.06]
  Week 16 (n=38,38,14,15) | -9.38 (1.927) [0.00 to 3.51] | -6.63 (1.936) [NA to NA] | 2.04 (3.151) [NA to NA] | 0.84 (3.082) [0.00 to 7.52]
  Week 20 (n=37,38,14,15) | -12.68 (1.886) [NA to NA] | -9.18 (1.884) [NA to NA] | 0.48 (3.079) [NA to NA] | 2.04 (2.999) [NA to NA]
  Week 32 (n=37,37,14,14) | -14.02 (2.350) [NA to NA] | -11.31 (2.350) [NA to NA] | -11.81 (3.834) [NA to NA] | -12.61 (3.788) [NA to NA]
  Week 40 (n=36,36,13,13) | -16.31 (2.365) [0.00 to 3.68] | -11.94 (2.359) [NA to NA] | -13.42 (3.876) [NA to NA] | -14.19 (3.842) [NA to NA]
  Week 52 (n=31,34,12,13) | -17.13 (2.689) | -13.55 (2.651) | -15.08 (4.387) | -17.89 (4.315)

31. Secondary Outcome: Number of Affected Nails in Participants With Nail Psoriasis at Baseline Over Time Through Week 52
Description: Nail psoriasis is evaluated by the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Total number psoriasis affected nails (presence of psoriatic manifestations on the nail matrix/nail bed) were assessed and reported. The total number of affected FINGER nails was reported.
Time Frame: Baseline and Weeks 8, 16, 20, 32, 40, and 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nails
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 40 | 38 | 18 | 18
nails
  Baseline (n=40,38,18,18) | 7.6 (3.06) [0.00 to 3.51] | 7.3 (3.21) [0.00 to 5.64] | 8.1 (2.97) [0.77 to 20.28] | 7.4 (3.45) [0.00 to 16.06]
  Week 8 (n=39,38,15,15) | 7.2 (3.07) [0.00 to 3.51] | 7.2 (3.61) [NA to NA] | 7.3 (3.58) [NA to NA] | 7.9 (3.20) [0.00 to 7.52]
  Week 16 (n=38,38,14,15) | 6.1 (3.53) [NA to NA] | 6.6 (3.57) [NA to NA] | 7.9 (3.82) [NA to NA] | 7.6 (3.56) [NA to NA]
  Week 20 (n=37,38,14,15) | 5.1 (3.84) [NA to NA] | 6.0 (3.84) [NA to NA] | 7.4 (3.93) [NA to NA] | 7.9 (3.08) [NA to NA]
  Week 32 (n=37,37,14,14) | 3.8 (3.92) [0.00 to 3.68] | 5.5 (3.85) [NA to NA] | 6.1 (3.95) [NA to NA] | 7.6 (3.72) [NA to NA]
  Week 40 (n=36,36,13,13) | 3.0 (3.60) | 5.4 (4.08) | 6.3 (4.39) | 5.8 (4.28)
  Week 52 (n=31,34,12,13) | 3.0 (3.67) | 4.4 (4.23) | 4.6 (4.12) | 4.4 (3.75)

32. Secondary Outcome: Percent Change From Baseline in NAPSI Over Time Through Week 52
Description: as for outcome 29
Time Frame: Baseline and weeks 8, 16, 20, 32, 40, and 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Tofacitinib 10 mg: Participants received tofacitinib 10 mg tablet orally twice daily (approximately 12 0hours apart) up to Week 52.
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 40 | 38 | 18 | 18
percent change
  Week 8 (n=39,38,15,15) | -9.59 (8.473) [0.00 to 3.51] | -8.81 (8.585) [NA to NA] | 5.28 (13.661) [NA to NA] | 25.40 (13.662) [0.00 to 7.52]
  Week 16 (n=38,38,14,15) | -33.31 (10.552) [NA to NA] | -14.91 (10.600) [NA to NA] | -3.26 (17.257) [NA to NA] | 18.43 (16.869) [NA to NA]
  Week 20 (n=37,38,14,15) | -51.97 (8.748) [NA to NA] | -25.10 (8.715) [NA to NA] | -8.87 (14.276) [NA to NA] | 13.72 (13.869) [NA to NA]
  Week 32 (n=37,37,14,14) | -58.44 (10.256) [0.00 to 3.68] | -25.27 (10.247) [NA to NA] | -50.20 (16.734) [NA to NA] | -45.83 (16.481) [NA to NA]
  Week 40 (n=36,36,13,13) | -68.68 (9.243) | -37.40 (9.208) | -47.17 (15.143) | -58.60 (14.988)
  Week 52 (n=31,34,12,13) | -71.40 (10.891) | -51.71 (10.636) | -56.08 (17.621) | -45.67 (17.192)

33. Secondary Outcome: Percentage of Participants With NAPSI75 Response Over Time Through Week 52
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores represents more severe psoriasis. NAPSI 75 response was defined as at least a 75% reduction in NAPSI relative to Baseline. Percentage of participants with NAPSI 75 response is reported.
Time Frame: Weeks 8, 16, 20, 32, 40, and 52
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 40 | 38 | 18 | 18
percentage of participants
  Week 8 | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 10.53 [0.77 to 20.28] | 5.56 [0.00 to 16.14] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 16 | 20.00 [7.60 to 32.40] | 15.79 [4.20 to 27.38] | 11.11 [0.00 to 25.63] | 5.56 [0.00 to 16.14]
  Week 20 | 30.00 [15.80 to 44.20] | 13.16 [2.41 to 23.91] | 11.11 [0.00 to 25.63] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 32 | 52.50 [37.02 to 67.98] | 28.95 [14.53 to 43.37] | 27.78 [7.09 to 48.47] | 16.67 [0.00 to 33.88]
  Week 40 | 65.00 [50.22 to 79.78] | 34.21 [19.13 to 49.29] | 33.33 [11.56 to 55.11] | 33.33 [11.56 to 55.11]
  Week 52 | 52.50 [37.02 to 67.98] | 47.37 [31.49 to 63.24] | 38.89 [16.37 to 61.41] | 38.89 [16.37 to 61.41]

34. Secondary Outcome: Percentage of Participants With NAPSI100 Response Over Time Through Week 52
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores represents more severe psoriasis. NAPSI 100 response was defined as at least a 100% reduction in NAPSI relative to Baseline. Percentage of participants with NAPSI 100 response is reported.
Time Frame: Weeks 8, 16, 20, 32, 40, and 52
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 40 | 38 | 18 | 18
percentage of participants
  Week 8 | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 5.26 [0.00 to 12.36] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 16 | 5.00 [0.00 to 11.75] | 5.26 [0.00 to 12.36] | 11.11 [0.00 to 25.63] | 5.56 [0.00 to 16.14]
  Week 20 | 17.50 [5.72 to 29.28] | 10.53 [0.77 to 20.28] | 11.11 [0.00 to 25.63] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 32 | 27.50 [13.66 to 41.34] | 13.16 [2.41 to 23.91] | 11.11 [0.00 to 25.63] | 5.56 [0.00 to 16.14]
  Week 40 | 30.00 [15.80 to 44.20] | 15.79 [4.20 to 27.38] | 11.11 [0.00 to 25.63] | 16.67 [0.00 to 33.88]
  Week 52 | 30.00 [15.80 to 44.20] | 31.58 [16.80 to 46.36] | 16.67 [0.00 to 33.88] | 16.67 [0.00 to 33.88]

35. Secondary Outcome: Actual Itch Severity Item (ISI) Score Over Time Through Week 52
Description: ISI assessed severity of itch (pruritus) due to psoriasis. ISI is a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends for post baseline time points. Baseline ISI is average of scores on 7 days prior to start of study treatment.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Baseline (n=88,88,44,44) | 5.66 (2.586) [NA to NA] | 5.10 (2.679) [0.00 to 12.36] | 5.22 (2.501) [NA to NA] | 5.75 (2.679) [NA to NA]
  Week 2 (n=87,86,44,42) | 2.97 (2.043) [0.00 to 11.75] | 3.49 (2.669) [0.00 to 12.36] | 5.45 (2.791) [0.00 to 25.63] | 4.95 (2.731) [0.00 to 16.14]
  Week 4 (n=88,88,43,42) | 2.13 (2.061) [5.72 to 29.28] | 2.68 (2.322) [0.77 to 20.28] | 5.23 (2.715) [0.00 to 25.63] | 5.12 (2.491) [NA to NA]
  Week 8 (n=85,88,40,39) | 1.47 (1.900) [13.66 to 41.34] | 2.41 (2.283) [2.41 to 23.91] | 4.75 (2.677) [0.00 to 25.63] | 4.97 (2.978) [0.00 to 16.14]
  Week 12 (n=84,88,40,39) | 1.24 (1.565) [15.80 to 44.20] | 2.13 (2.323) [4.20 to 27.38] | 4.00 (2.621) [0.00 to 25.63] | 5.00 (2.938) [0.00 to 33.88]
  Week 16 (n=84,84,38,39) | 1.17 (1.782) [15.80 to 44.20] | 2.01 (2.367) [16.80 to 46.36] | 3.89 (2.391) [0.00 to 33.88] | 5.13 (2.811) [0.00 to 33.88]
  Week 20 (n=83,84,38,38) | 1.06 (1.564) | 2.01 (2.326) | 1.95 (2.253) | 2.11 (2.227)
  Week 32 (n=838238,37 | 0.88 (1.273) | 2.07 (2.382) | 1.24 (1.747) | 1.51 (2.388)
  Week 40 (n=81,81,37,36) | 0.96 (1.145) | 2.30 (2.283) | 1.49 (2.181) | 1.53 (2.158)
  Week 52 (n=80,78,36,36) | 1.45 (2.074) | 2.55 (2.516) | 1.89 (2.482) | 2.36 (2.380)

36. Secondary Outcome: Change From Baseline in ISI Score Over Time Through Week 52
Description: ISI assessed severity of itch (pruritus) due to psoriasis. ISI is a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends.
Time Frame: Baseline and weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Week 2 (n=86,86,44,42) | -2.50 (0.219) [0.00 to 11.75] | -1.76 (0.218) [0.00 to 12.36] | 0.12 (0.306) [0.00 to 25.63] | -0.64 (0.314) [0.00 to 16.14]
  Week 4 (n=87,88,43,42) | -3.33 (0.226) [5.72 to 29.28] | -2.60 (0.224) [0.77 to 20.28] | -0.03 (0.319) [0.00 to 25.63] | -0.47 (0.325) [NA to NA]
  Week 8 (n=84,88,40,39) | -3.93 (0.232) [13.66 to 41.34] | -2.88 (0.228) [2.41 to 23.91] | -0.50 (0.331) [0.00 to 25.63] | -0.46 (0.337) [0.00 to 16.14]
  Week 12 (n=83,88,40,39) | -4.10 (0.237) [15.80 to 44.20] | -3.16 (0.233) [4.20 to 27.38] | -1.15 (0.338) [0.00 to 25.63] | -0.44 (0.344) [0.00 to 33.88]
  Week 16 (n=83,84,38,39) | -4.21 (0.232) [15.80 to 44.20] | -3.28 (0.229) [16.80 to 46.36] | -1.30 (0.335) [0.00 to 33.88] | -0.33 (0.337) [0.00 to 33.88]
  Week 20 (n=82,84,38,38) | -4.32 (0.219) | -3.28 (0.216) | -3.22 (0.318) | -3.36 (0.320)
  Week 32 (n=82,82,38,37) | -4.51 (0.220) | -3.17 (0.219) | -4.01 (0.322) | -4.04 (0.325)
  Week 40 (n=80,81,37,36) | -4.39 (0.224) | -2.98 (0.222) | -3.81 (0.328) | -3.89 (0.331)
  Week 52 (n=79,78,36,36) | -3.91 (0.272) | -2.71 (0.272) | -3.47 (0.401) | -3.11 (0.403)

37. Secondary Outcome: Actual Dermatology Life Quality Index (DLQI) Score Over Time Through Week 52
Description: as for outcome 5
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Baseline (n=90,88,44,44) | 14.1 (7.17) [0.00 to 11.75] | 13.5 (7.29) [0.00 to 12.36] | 12.5 (6.82) [0.00 to 25.63] | 12.1 (6.92) [0.00 to 16.14]
  Week 2 (n=88,86,44,42) | 9.5 (5.31) [5.72 to 29.28] | 10.0 (6.20) [0.77 to 20.28] | 12.6 (7.34) [0.00 to 25.63] | 10.4 (5.97) [NA to NA]
  Week 4 (n=86,88,42,41) | 7.6 (5.00) [13.66 to 41.34] | 8.2 (5.46) [2.41 to 23.91] | 12.4 (7.99) [0.00 to 25.63] | 10.3 (5.39) [0.00 to 16.14]
  Week 8 (n=85,88,40,39) | 5.9 (5.49) [15.80 to 44.20] | 7.5 (5.89) [4.20 to 27.38] | 11.2 (7.25) [0.00 to 25.63] | 9.9 (6.66) [0.00 to 33.88]
  Week 12 (n=84,88,39,39) | 4.6 (4.47) [15.80 to 44.20] | 6.7 (6.16) [16.80 to 46.36] | 11.1 (7.11) [0.00 to 33.88] | 10.2 (6.86) [0.00 to 33.88]
  Week 16 (n=84,84,38,39) | 4.3 (4.70) | 6.2 (5.62) | 10.7 (7.20) | 10.5 (6.77)
  Week 20 (n=82,84,38,39) | 3.8 (4.46) | 5.4 (5.50) | 6.2 (4.80) | 6.4 (5.17)
  Week 32 (n=83,82,38,37) | 3.2 (4.39) | 5.1 (5.31) | 4.7 (5.42) | 5.0 (6.03)
  Week 40 (n=81,81,37,36) | 3.7 (4.37) | 5.9 (5.44) | 4.6 (5.07) | 4.1 (4.03)
  Week 52 (n=80,78,35,36) | 4.6 (5.83) | 6.5 (6.25) | 4.7 (5.85) | 6.0 (5.68)

38. Secondary Outcome: Change From Baseline in DLQI Score Over Time Through Week 52
Description: as for outcome 5
Time Frame: Baseline and weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Week 2 (n=88,86,44,42) | -3.98 (0.455) [0.00 to 11.75] | -3.26 (0.458) [0.00 to 12.36] | -0.20 (0.644) [0.00 to 25.63] | -2.27 (0.659) [0.00 to 16.14]
  Week 4 (n=86,88,44,42) | -5.96 (0.492) [5.72 to 29.28] | -5.11 (0.488) [0.77 to 20.28] | 0.17 (0.700) [0.00 to 25.63] | -2.26 (0.712) [NA to NA]
  Week 8 (n=85,88,40,39) | -7.52 (0.594) [13.66 to 41.34] | -5.83 (0.587) [2.41 to 23.91] | -1.00 (0.852) [0.00 to 25.63] | -2.70 (0.868) [0.00 to 16.14]
  Week 12 (n=84,88,39,39) | -8.59 (0.618) [15.80 to 44.20] | -6.64 (0.609) [4.20 to 27.38] | -0.76 (0.891) [0.00 to 25.63] | -2.44 (0.904) [0.00 to 33.88]
  Week 16 (n=84,84,38,39) | -9.03 (0.618) [15.80 to 44.20] | -7.00 (0.611) [16.80 to 46.36] | -1.15 (0.899) [0.00 to 33.88] | -2.22 (0.905) [0.00 to 33.88]
  Week 20 (n=82,84,38,39) | -9.36 (0.562) | -7.78 (0.555) | -5.84 (0.819) | -6.30 (0.821)
  Week 32 (n=83,82,38,37) | -10.05 (0.565) | -8.07 (0.562) | -7.44 (0.828) | -7.94 (0.837)
  Week 40 (n=81,81,37,36) | -9.56 (0.563) | -7.32 (0.559) | -7.61 (0.826) | -8.28 (0.836)
  Week 52 (n=80,78,35,36) | -8.63 (0.679) | -6.63 (0.681) | -7.42 (1.012) | -6.37 (1.010)

39. Secondary Outcome: Percentage of Participants With Patient Global Assessment (PtGA) Response of "Clear" or "Almost Clear" Over Time Through Week 52
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5-point scale (0=clear [no psoriasis]; 1=almost clear; 2=mild; 3=moderate; 4=severe). the percentage of participants with scores of 0 (clear) and 1 (almost clear) are reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
percentage of participants
  Week 2 | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's. | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 4 | 7.78 [2.24 to 13.31] | 5.68 [0.85 to 10.52] | 2.27 [0.00 to 6.68] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 8 | 32.22 [22.57 to 41.88] | 19.32 [11.07 to 27.57] | 2.27 [0.00 to 6.68] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 12 | 45.56 [35.27 to 55.84] | 27.27 [17.97 to 36.58] | 2.27 [0.00 to 6.68] | 0.00 [NA to NA] — It is because the calculation method is based on normal approximation which assumes a big sample size, but n=0 at these weeks. Hence, it's not appropriate to use normal approximation to estimate the CI's.
  Week 16 | 55.56 [45.29 to 65.82] | 34.09 [24.19 to 43.99] | 9.09 [0.60 to 17.59] | 4.55 [0.00 to 10.70]
  Week 20 | 52.22 [41.90 to 62.54] | 31.82 [22.09 to 41.55] | 18.18 [6.79 to 29.58] | 13.64 [3.50 to 23.78]
  Week 32 | 56.67 [46.43 to 66.90] | 34.09 [24.19 to 43.99] | 45.45 [30.74 to 60.17] | 31.82 [18.06 to 45.58]
  Week 40 | 52.22 [41.90 to 62.54] | 34.09 [24.19 to 43.99] | 50.00 [35.23 to 64.77] | 40.91 [26.38 to 55.44]
  Week 52 | 51.11 [40.78 to 61.44] | 26.14 [16.96 to 35.32] | 47.73 [32.97 to 62.49] | 29.55 [16.06 to 43.03]

40. Secondary Outcome: Euro Quality of Life 5 Dimensions (EQ-5D) - Utility Score Over Time Through Week 52
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a worse health state.
Time Frame: Baseline, Weeks 16, 32, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Baseline (n=90,88,44,44) | 0.784 (0.2088) [NA to NA] | 0.797 (0.1991) [NA to NA] | 0.779 (0.1803) [NA to NA] | 0.741 (0.2183) [NA to NA]
  Week 16 (n=84,83,38,39) | 0.957 (0.0778) [2.24 to 13.31] | 0.930 (0.1226) [0.85 to 10.52] | 0.905 (0.1191) [0.00 to 6.68] | 0.817 (0.2108) [NA to NA]
  Week 32 (n=83,82,38,37) | 0.955 (0.0796) [22.57 to 41.88] | 0.904 (0.1368) [11.07 to 27.57] | 0.960 (0.0739) [0.00 to 6.68] | 0.917 (0.1477) [NA to NA]
  Week 40 (n=81,81,37,36) | 0.950 (0.0940) [35.27 to 55.84] | 0.918 (0.1177) [17.97 to 36.58] | 0.954 (0.0776) [0.00 to 6.68] | 0.938 (0.1125) [NA to NA]
  Week 52 (n=80,78,35,36) | 0.938 (0.1303) [45.29 to 65.82] | 0.893 (0.1719) [24.19 to 43.99] | 0.941 (0.1118) [0.60 to 17.59] | 0.887 (0.1626) [0.00 to 10.70]

41. Secondary Outcome: Change From Baseline in EQ-5D - Utility Score Over Time Through Week 52
Description: as for outcome 40
Time Frame: Baseline and weeks 16, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Week 16 (n=84,83,38,39) | 0.172 (0.2164) [2.24 to 13.31] | 0.128 (0.2108) [0.85 to 10.52] | 0.105 (0.1824) [0.00 to 6.68] | 0.074 (0.2391) [NA to NA]
  Week 32 (n=83,82,38,37) | 0.170 (0.2092) [22.57 to 41.88] | 0.109 (0.2347) [11.07 to 27.57] | 0.160 (0.1904) [0.00 to 6.68] | 0.173 (0.2202) [NA to NA]
  Week 40 (n=81,81,37,36) | 0.168 (0.2159) [35.27 to 55.84] | 0.120 (0.2322) [17.97 to 36.58] | 0.159 (0.1937) [0.00 to 6.68] | 0.192 (0.2103) [NA to NA]
  Week 52 (n=80,78,35,36) | 0.156 (0.2071) [45.29 to 65.82] | 0.101 (0.2477) [24.19 to 43.99] | 0.147 (0.2136) [0.60 to 17.59] | 0.142 (0.2328) [0.00 to 10.70]

42. Secondary Outcome: Euro Quality of Life 5 Dimensions (EQ-5D) - Visual Analog Scale (VAS) Over Time Through Week 52
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeter (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline and Weeks 16, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Baseline (n=90,88,44,44) | 65.8 (24.90) [NA to NA] | 69.5 (19.84) [NA to NA] | 66.4 (23.09) [NA to NA] | 67.4 (21.92) [NA to NA]
  Week 16 (n=84,83,38,39) | 83.7 (15.30) [2.24 to 13.31] | 78.9 (15.41) [0.85 to 10.52] | 72.3 (22.04) [0.00 to 6.68] | 68.4 (20.20) [NA to NA]
  Week 32 (n=83,82,38,37) | 84.5 (16.17) [22.57 to 41.88] | 82.4 (16.00) [11.07 to 27.57] | 85.2 (14.36) [0.00 to 6.68] | 81.7 (17.25) [NA to NA]
  Week 40 (n=81,81,37,36) | 85.5 (14.45) [35.27 to 55.84] | 83.0 (14.35) [17.97 to 36.58] | 83.5 (16.86) [0.00 to 6.68] | 81.9 (16.03) [NA to NA]
  Week 52 (n=80,78,35,36) | 82.5 (17.13) [45.29 to 65.82] | 80.0 (18.40) [24.19 to 43.99] | 85.0 (13.58) [0.60 to 17.59] | 80.7 (19.20) [0.00 to 10.70]

43. Secondary Outcome: Change From Baseline in EQ-5D - Visual Analog Scale (VAS) Over Time Through Week 52
Description: as for outcome 42
Time Frame: Baseline and weeks 16, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
units on a scale
  Week 16 (n=84,83,38,39) | 17.5 (25.23) [2.24 to 13.31] | 8.8 (21.15) [0.85 to 10.52] | 2.6 (22.17) [0.00 to 6.68] | -0.6 (21.16)
  Week 32 (n=83,82,38,37) | 18.4 (25.92) | 13.1 (22.36) | 15.4 (23.50) | 12.2 (23.99)
  Week 40 (n=81,81,37,36) | 19.9 (27.07) | 13.3 (22.31) | 14.3 (23.19) | 11.8 (24.46)
  Week 52 (n=80,78,35,36) | 16.1 (26.08) | 9.9 (24.54) | 15.2 (22.96) | 10.7 (21.16)

44. Other Pre Specified Outcome: Treatment-Emergent All Causalities Adverse Events (AEs) During Week 0-16
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline to Week 16
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
participants
  Number of Participants with AEs(All Causalities) | 61 | 57 | 43
  Number of Participants with SAEs(All Causalities) | 0 | 2 | 0
  Number of Participants Discontinued due to AEs | 1 | 3 | 3

45. Other Pre Specified Outcome: Treatment-Emergent All Causalities Adverse Events (AEs) During Week 0-52
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline to Week 52
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
participants
  Number of Participants with AEs (All Causalities) | 76 | 74 | 35 | 33
  Number of Participants with SAEs(All Causalities) | 2 | 4 | 1 | 0
  Number of Participants Discontinued due to AEs | 1 | 3 | 3 | 1

46. Other Pre Specified Outcome: Number of Participants With Laboratory Values Meeting Protocol Criteria for Discontinuation During Week 0-16
Description: Study drugs were to be discontinued and the participant withdrawn for: 2 sequential absolute neutrophil counts (ANC) <1.0 X 10^9/L (1000/mm^3); 2 sequential absolute lymphocyte counts <0.5 X 10^9/L; 2 sequential hemoglobin values <9.0 g/dL and/or decreases of >30% from baseline value; 2 sequential platelet counts <75 X 10^9/L; 2 sequential AST or ALT elevations ≥3X ULN with at least 1 total bilirubin value ≥2X ULN (reason #1); 2 sequential AST or ALT elevations ≥5X ULN regardless of total bilirubin or accompanying signs or symptoms (reason #2); 2 sequential increases in serum creatinine >50% and an increase in serum creatinine >0.5 mg/dL over the average of screening and baseline values; 2 sequential CK elevations >10X ULN.
Time Frame: Baseline to Week 16
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
participants
  2 Sequential absolute neutrophil count | 0 | 0 | 0
  2 Sequential absolute lymphocyte count | 0 | 0 | 0
  2 Sequential hemoglobin | 0 | 0 | 0
  2 Sequential platelet count | 2 | 0 | 0
  2 Sequential AST or ALT reason #1 | 0 | 0 | 0
  2 Sequential AST or ALT reason #2 | 0 | 0 | 0
  2 Sequential serum creatinine | 0 | 0 | 0
  2 sequential creatine kinase | 0 | 0 | 0

47. Other Pre Specified Outcome: Number of Participants With Laboratory Values Meeting Protocol Criteria for Discontinuation During Week 0-52
Description: as for outcome 46
Time Frame: Baseline up to Week 52
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
participants
  2 Sequential absolute neutrophil count | 0 | 0 | 0 | 0
  2 Sequential absolute lymphocyte count | 0 | 0 | 0 | 0
  2 Sequential hemoglobin | 1 | 0 | 0 | 0
  2 Sequential platelet count | 2 | 0 | 0 | 1
  2 Sequential AST or ALT reason #1 | 0 | 0 | 0 | 0
  2 Sequential AST or ALT reason #2 | 0 | 1 | 0 | 0
  2 Sequential serum creatinine | 0 | 0 | 0 | 0
  2 sequential creatine kinase | 0 | 0 | 0 | 0

48. Other Pre Specified Outcome: Number of Participants With Vital Sign Values Meeting the Criteria for Potential Clinical Concern During Week 0-16
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: pulse rate less than (<)40 or greater than (>)120 beats per minute (bpm), heart rate less than (<)40 or greater than (>)120 bpm; sitting systolic blood pressure (SBP) of greater than or equal to (>=)30 millimeters of mercury (mmHg) change from baseline or sitting SBP <90 mmHg, sitting diastolic blood pressure (DBP) >=20 mmHg change from baseline or sitting DBP <50 mmHg.
Time Frame: Baseline to Week 16
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo; n=number of participants evaluated against criteria.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
participants
  Sitting SBP <90 mmHg (n=87,88,86) | 1 | 0 | 0
  Sitting DBP <50 mmHg (n=87,88,86) | 0 | 0 | 1
  Heart Rate <40 or >120 bpm (n=73,74,68) | 0 | 0 | 0
  Pulse Rate <40 or >120 bpm (n=84,85,82) | 0 | 0 | 0
  Sitting SBP max Increase >=30 Hg(n=87,88,86) | 1 | 0 | 0
  Sitting DBP max Increase >=20 mmHg(n=87,88,86) | 0 | 1 | 1
  Sitting SBP max Decrease >=30 mmHg(n=87,88,86) | 3 | 2 | 2
  Sitting DBP max Decrease >=20 mmHg(n=87,88,86) | 2 | 5 | 1

49. Other Pre Specified Outcome: Number of Participants With Vital Sign Values Meeting the Criteria for Potential Clinical Concern During Week 0-52
Description: as for outcome 48
Time Frame: Baseline to Week 52
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo; n=number of evaluable participants at the specified time point.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
participants
  Sitting SBP <90 mmHg (n=87,88,44,42) | 1 | 0 | 0 | 0
  Sitting DBP <50 mmHg (n=87,88,44,42) | 0 | 0 | 0 | 1
  Heart Rate <40 or >120 bpm (n=74,75,35,34) | 0 | 0 | 0 | 0
  Pulse Rate <40 or >120 bpm (n=86,85,42,40) | 0 | 0 | 0 | 0
  Sitting SBP max Increase >=30 Hg(n=87,88,44,42) | 5 | 1 | 1 | 2
  Sitting DBP max Increase >=20 mmHg(n=87,88,44,42) | 5 | 4 | 2 | 1
  Sitting SBP max Decrease >=30 mmHg(n=87,88,44,42) | 4 | 3 | 2 | 1
  Sitting DBP max Decrease >=20 mmHg(n=87,88,44,42) | 3 | 8 | 1 | 1

50. Other Pre Specified Outcome: Incidence of Participants With Adjudicated Cardiovascular (CV) Endpoints Reported During Week 0-16
Description: CV event categories included: cerebrovascular accident (CVA), coronary revascularization procedure (percutaneous transluminal coronary angioplasty [PTCA], percutaneous coronary intervention [PCI], coronary bypass grafting [CABG], heart failure, major adverse cardiac events (MACE), myocardial infarction (MI), new ischemic heart disease, peripheral vascular disease (first diagnosis). MACE included any MI, CVA (stroke or transient ischemic attack), or CV death.
Time Frame: Baseline to Week 16
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
participants
  Cerebrovascular Accident | 0 | 0 | 0
  Coronary Revascularization Procedure | 0 | 0 | 0
  Heart Failure | 0 | 0 | 0
  MACE | 0 | 0 | 0
  Myocardial Infarction | 0 | 0 | 0
  New Ischemic Heart Disease | 0 | 0 | 0
  Peripheral Vascular Disease | 0 | 0 | 0
  Non-CV Death | 0 | 1 | 0

51. Other Pre Specified Outcome: Incidence of Participants With Adjudicated Cardiovascular (CV) Endpoints Reported During Week 0-52
Description: as for outcome 50
Time Frame: Baseline up to Week 52
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
participants
  Cerebrovascular Accident | 0 | 0 | 0 | 0
  Coronary Revascularization Procedure | 0 | 1 | 1 | 0
  Heart Failure | 0 | 0 | 0 | 0
  MACE | 0 | 0 | 0 | 0
  Myocardial Infarction | 0 | 0 | 0 | 0
  New Ischemic Heart Disease | 0 | 0 | 0 | 0
  Peripheral Vascular Disease | 0 | 0 | 0 | 0
  Non-CV Death | 0 | 1 | 0 | 0

52. Other Pre Specified Outcome: Number of Participants With Adjudicated Malignancy Events Reported During Week 0-16
Description: As part of AE monitoring, potential malignancy events were adjudicated and centrally reviewed by a safety committee.
Time Frame: Baseline to Week 16
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo
Number analyzed (Participants) | 90 | 88 | 88
participants | 0 | 1 | 0

53. Other Pre Specified Outcome: Number of Participants With Adjudicated Malignancy Events Reported During Week 0-52
Description: As part of AE monitoring, potential malignancy events were adjudicated and centrally reviewed by a safety committee.
Time Frame: Baseline to Week 52
Population: The safety analysis set included all participants who received at least 1 dose of tofacitinib or placebo.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg
Number analyzed (Participants) | 90 | 88 | 44 | 44
participants | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and a non-serious event during the study.
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg | Placebo to Tofacitinib 10 mg | Placebo to Tofacitinib 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/90 | 4/88 | 1/44 | 0/44 | 0/88
Other Adverse Events (participants affected / at risk) | 59/90 | 60/88 | 25/44 | 31/44 | 23/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg (N=90) | Tofacitinib 5 mg (N=88) | Placebo to Tofacitinib 10 mg (N=44) | Placebo to Tofacitinib 5 mg (N=44) | Placebo (N=88)
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tofacitinib 10 mg (N=90) | Tofacitinib 5 mg (N=88) | Placebo to Tofacitinib 10 mg (N=44) | Placebo to Tofacitinib 5 mg (N=44) | Placebo (N=88)
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 11 | 12 | 6 | 9 | 3
Upper respiratory tract infection (Infections and infestations) | 11 | 18 | 5 | 7 | 3
Blood cholesterol increased (Investigations) | 15 | 9 | 1 | 3 | 2
Blood triglycerides increased (Investigations) | 8 | 11 | 4 | 2 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 15 | 13 | 8 | 7 | 9
Hypomenorrhoea (Reproductive system and breast disorders) | 0/23 | 2/23 | 0/14 | 0/12 | 0/26 — This event is limited to female participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 5 | 5 | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 5 | 1 | 3 | 3 | 5
Toothache (Gastrointestinal disorders) | 5 | 1 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 5 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 5 | 3 | 2 | 1 | 0
Influenza (Infections and infestations) | 2 | 2 | 1 | 3 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/23 | 1/23 | 1/14 | 0/12 | 0/26 — This event is limited to female participants.
Alanine aminotransferase increased (Investigations) | 9 | 4 | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 0 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 5 | 1 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 5 | 4 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 6 | 2 | 1 | 1 | 0
Low density lipoprotein increased (Investigations) | 8 | 6 | 0 | 2 | 0
Protein urine present (Investigations) | 5 | 4 | 3 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1/23 | 2/23 | 0/14 | 1/12 | 0/26 — This event is limited to female participants.
Vulvovaginal candidiasis (Infections and infestations) | 0/23 | 0/23 | 0/14 | 1/12 | 0/26 — This event is limited to female participants.
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.